

### CLINICAL STUDY PROTOCOL

Study Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study

Evaluating the Safety, Tolerability, and Efficacy of GS-9674 in

Subjects with Nonalcoholic Steatohepatitis (NASH)

Sponsor: Gilead Sciences, Inc.

333 Lakeside Drive Foster City, CA 94404

U.S.A.

**IND Number:** 127960

EudraCT Number: 2016-002496-10 Clinical Trials.gov NCT02854605

Identifier:

Indication: Nonalcoholic steatohepatitis (NASH)

Protocol ID: GS-US-402-1852

Gilead Medical Name: C. Stephen Djedjos, M.D.

Monitor: Telephone: PPD

Fax: PPD Email: PPD

Protocol Version/Date: Original: 28 June 2016

Amendment 1: 03-October-2016

### CONFIDENTIALITY STATEMENT

The information contained in this document, particularly unpublished data, is the property or under control of Gilead Sciences, Inc., and is provided to you in confidence as an investigator, potential investigator, or consultant, for review by you, your staff, and an applicable Institutional Review Board or Independent Ethics Committee. The information is only to be used by you in connection with authorized clinical studies of the investigational drug described in the protocol. You will not disclose any of the information to others without written authorization from Gilead Sciences, Inc., except to the extent necessary to obtain informed consent from those persons to whom the drug may be administered.

# **TABLE OF CONTENTS**

| TABL | LE OF CONTENTS | 2 |
|---|---|---|
| LIST | OF IN-TEXT TABLES | 5 |
| LIST | OF IN-TEXT FIGURES | 5 |
| PROT | TOCOL SYNOPSIS | 6 |
| | SSARY OF ABBREVIATIONS AND DEFINITION OF TERMS | |
| 1. I | INTRODUCTION | |
| 1 | 1.1. Background | |
| | 1.1.1. GS-9674 General Information | |
| | 1.1.2. Nonclinical Toxicology | |
| | 1.1.4. Nonclinical Pharmacokinetics | |
| | 1.1.5. Clinical Trials of GS-9674 | |
| 1 | 1.2. Rationale for This Study | |
| | 1.3. Risk/Benefit Assessment for the Study | |
| 1 | 1.4. Compliance | |
| 2. ( | OBJECTIVES | 27 |
| | STUDY DESIGN | |
| | 3.1. Study Design | |
| | 3.2. Treatment Plan and Regimen | |
| 3 | 3.3. Biomarker Testing | |
| | 3.3.1. Biomarker Samples to Address the Study Objectives | |
| | <ul><li>3.3.2. Biomarker Samples for Optional Future Research</li><li>3.3.3. Biomarker Samples for Optional Genomic Research</li></ul> | |
| 4. § | SUBJECT POPULATION | |
| | 4.1. Number of Subjects and Subject Selection | |
| | 4.2. Inclusion Criteria | |
| 4 | 4.3. Exclusion Criteria | 32 |
| 5. I | INVESTIGATIONAL MEDICINAL PRODUCTS | 35 |
| 5 | 5.1. Randomization, Blinding and Treatment Codes | 35 |
| | 5.1.1. Procedures for Breaking Treatment Codes | 35 |
| 5 | 5.2. Description and Handling of GS-9674 and PTM GS-9674 | 36 |
| | 5.2.1. Formulation | |
| | 5.2.2. Packaging and Labeling | |
| _ | 5.2.3. Storage and Handling | |
| | 5.3. Dosage and Administration of GS-9674/ PTM GS-9674 | |
| | 5.4. Prior and Concomitant Medications | |
| | <ul><li>5.5. Prohibited Medications</li><li>5.6. Accountability for GS-9674/ PTM GS-9674</li></ul> | |
| - | 5.6.1. Investigational Medicinal Product Return or Disposal | |
| | - | |
| | STUDY PROCEDURES | |
| | 6.1. Subject Enrollment and Treatment Assignment | |
| | 6.2. Pretreatment Assessments – Screening Visit | |
| | 6.3. Baseline/Day 1 Randomization and Assessments | |
| ( | U.T. I TORUMONI (ASSUSSIMENTS) | 43 |

| | | 6.4.1. Week 1 | 43 |
|---|---|---|---|
| | | 6.4.2. Week 4 Visit | |
| | | 6.4.3. Week 8, 16, and 20 Visits | |
| | | 6.4.4. Week 12 Visit | 46 |
| | | 6.4.5. Week 24 Visit | |
| | | 6.4.6. Unscheduled Visits. | |
| | 6.5. | Follow-Up Visit | 49 |
| | 6.6. | Assessments for Premature Discontinuation from Study | 49 |
| | 6.7. | Criteria for Discontinuation of Study Treatment. | 50 |
| | 6.8. | PK and PD Substudy Visits | 50 |
| | 6.9. | Description of Assessments | 51 |
| | | 6.9.1. Clinical Laboratory Analytes | 51 |
| | | 6.9.2. Medical History | 52 |
| | | 6.9.3. Physical Examination | 52 |
| | | 6.9.4. Quality of Life (QoL) Assessments | 52 |
| | | 6.9.5. Electrocardiogram | 53 |
| | | 6.9.6. FibroScan <sup>®</sup> | 53 |
| | | 6.9.7. MRE and MRI-PDFF | 53 |
| | 6.10. | End of Study Definition | 54 |
| | 6.11. | Post Study Care | 54 |
| 7. | ADVE | ERSE EVENTS AND TOXICITY MANAGEMENT | 55 |
| | 7.1. | Definitions of Adverse Events, Adverse Reactions, and Serious Adverse Events | |
| | 7.1. | 7.1.1. Adverse Events | 55 |
| | | 7.1.2. Serious Adverse Events | |
| | | | 33 |
| | | 7.1.3. Clinical Laboratory Abnormalities and Other Abnormal Assessments as Adverse Events or Serious Adverse Events | 56 |
| | 7.2 | | |
| | 7.2. | Assessment of Adverse Events and Serious Adverse Events | |
| | | 7.2.1. Assessment of Causality for Study Drugs and Procedures | |
| | 7.2 | 7.2.2. Assessment of Severity | |
| | 7.3. | Investigator Requirements and Instructions for Reporting Adverse Events and Serious | 57 |
| | 7.4 | Adverse Events to Gilead | |
| | 7.4. | Gilead Reporting Requirements | |
| | 7.5. | Toxicity Management | |
| | 7.6. | Special Situations Reports. | |
| | | 7.6.1. Definitions of Special Situations | |
| | | 7.6.2. Instructions for Reporting Special Situations | |
| 8. | STAT | ISTICAL CONSIDERATIONS | 65 |
| | 8.1. | Analysis Objectives and Endpoints | 65 |
| | | 8.1.1. Analysis Objectives | 65 |
| | | 8.1.2. Primary Endpoint | 65 |
| | | 8.1.3. Exploratory Efficacy Endpoints | 66 |
| | 8.2. | Analysis Conventions. | 66 |
| | | 8.2.1. Analysis Sets | 66 |
| | | 8.2.2. Interim Analysis | 68 |
| | 8.3. | Data Handling Conventions | |
| | 8.4. | Demographic Data and Baseline Characteristics | 68 |
| | 8.5. | Efficacy Analysis | 68 |
| | 8.6. | Safety Analysis. | 69 |
| | | 8.6.1. Extent of Exposure | 69 |
| | | 8.6.2. Adverse Events | 69 |
| | | 8.6.3. Laboratory Evaluations | |
| | | 8.6.4. Other Safety Evaluations | 70 |

| | 8.7. | Pharmac | cokinetic Analysis | 70 |
|---|---|---|---|---|
| | 8.8. | | codynamic Analysis | |
| | 8.9. | | ker Analysis | |
| | 8.10. | Sample | Size | 70 |
| | 8.11. | Data Mo | onitoring Committee | 71 |
| 9. | RESP | ONSIBIL | ITIES | 72 |
| | 9.1. | Investig | ator Responsibilities | 72 |
| | | 9.1.1. | Good Clinical Practice | |
| | | 9.1.2. | Institutional Review Board (IRB)/Independent Ethics Committee (IEC)/ | |
| | | | Ethics Committee (EC) Review and Approval | 72 |
| | | 9.1.3. | Informed Consent | |
| | | 9.1.4. | Confidentiality | 73 |
| | | 9.1.5. | Study Files and Retention of Records | 73 |
| | | 9.1.6. | Case Report Forms | 74 |
| | | 9.1.7. | Investigational Medicinal Product Accountability and Return | 75 |
| | | 9.1.8. | Inspections | 75 |
| | | 9.1.9. | Protocol Compliance | |
| | 9.2. | Sponsor | Responsibilities | 76 |
| | | 9.2.1. | Protocol Modifications | 76 |
| | | 9.2.2. | Study Report and Publications | 76 |
| | 9.3. | Joint Inv | vestigator/Sponsor Responsibilities | 76 |
| | | 9.3.1. | Payment Reporting | 76 |
| | | 9.3.2. | Access to Information for Monitoring | 77 |
| | | 9.3.3. | Monitoring and Oversight of Biomarker Specimens | 77 |
| | | 9.3.4. | Access to Information for Auditing or Inspections | 77 |
| | | 9.3.5. | Study Discontinuation | 77 |
| 10. | REFE | RENCES | | 78 |
| 11. | APPE | NDICES . | | 81 |
| | Apper | ıdix 1. | Investigator Signature Page | 82 |
| | Appendix 2. | | Study Procedures Table for GS-US-402-1852 | |
| | Appendix 3. | | CTCAE Grading Scale for Severity of Adverse Events and Laboratory | 0.5 |
| | Appen | idix 4. | Abnormalities | 87 |
| | rippondix i. | | Contracentive Requirements | 88 |

# LIST OF IN-TEXT TABLES

| Table 1-1. | Exposure Margins for GS-9674 Based on Observed GS-9674 Exposure After Administration of 100 mg GS-9674 Under Fed Conditions in Cohort 5 Compared to Exposures Observed at NOAEL Doses in Mouse and Cynomolgus Monkey | 18 |
|---|---|---|
| Table 1-2. | Preliminary Pharmacokinetic Results from Study GS-US-402-2102 Evaluating the | |
| Table 1-3. | Effect of DDIs on Administration of 100 mg GS-9674 with Food (Cohorts 1-3) | 22 |
| | OATP/BCRP (Cohorts 5-6) | 23 |
| Table 5-1. | List of Medications Prohibited and to be used with Caution | 38 |
| | LIST OF IN-TEXT FIGURES | |
| Figure 3-1. | Overall Study Design | 28 |

### PROTOCOL SYNOPSIS

Gilead Sciences, Inc. 333 Lakeside Dr. Foster City, CA 94404, U.S.A.

| C4 1 TP41 | A DI 2 D 1 1 D 11 DI 1 D 1 C 4 11 1 C | G 1 |
|---|---|---|
| Study Title: | A Phase 2. Randomized, Double-Blind, Placebo-Controlled S | Mildv |

Evaluating the Safety, Tolerability, and Efficacy of GS-9674 in Subjects

with Nonalcoholic Steatohepatitis (NASH)

IND Number: EudraCT Number:

127960

Clinical Trials.gov Identifier: 2016-002496-10

NCT02854605

**Study Centers Planned:** 

Approximately 50 centers in North America, Europe, and Asia Pacific

**Objectives:** 

The primary objective of this study is to evaluate the safety and tolerability of GS-9674 in subjects with NASH as assessed by magnetic resonance imaging-proton density fat fraction (MRI-PDFF) and magnetic resonance elastography (MRE).

The exploratory objectives of this study are listed in Section 2.

**Study Design:** 

This is a Phase 2, randomized, double-blind, placebo-controlled study evaluating the safety, tolerability, and efficacy of GS-9674 in subjects with NASH as assessed by MRI-PDFF and MRE.

Participation in the study can last up to 32 weeks, which includes a 4-week screening period, a 24-week treatment period during which study drug will be administered, and a 4-week follow-up period. The screening period may be extended under special circumstances with the explicit approval of the Medical Monitor.

Subjects meeting the study's entry criteria will be randomly assigned in a 2:2:1 ratio to 1 of 3 treatment groups as shown in the figure below:



Randomization will be stratified by the presence or absence of diabetes mellitus as determined by medical history, use of medication for indication of diabetes mellitus, or based on screening lab values if previously undiagnosed (ie, hemoglobin A1c  $\geq$  6.5% OR fasting plasma glucose  $\geq 126 \text{ mg/dL}$ ).

| Num | ber o | f Su | bjects |
|-----|-------|------|--------|
| | Plan | ned: | |

Approximately 125 Subjects

Target Population:

Males and non-pregnant females between 18-75 years of age without cirrhosis and with NASH as assessed by magnetic resonance imaging (MRI) and magnetic resonance elastography (MRE).

Duration of Treatment:

24 Weeks

Diagnosis and Main Eligibility Criteria:

Key inclusion and exclusion criteria are as follows:

### **Inclusion Criteria:**

- Meets all of the following conditions:
  - a. A clinical diagnosis of nonalcoholic fatty liver disease (NAFLD) with histological or imaging evidence of fatty liver within the past two years. If necessary an ultrasound may be performed during screening to confirm NAFLD. Note: criterion a. must be met before evaluating criteria b. and c.
  - b. Screening MRI-PDFF with  $\geq 10\%$  steatosis
  - c. Screening MRE with liver stiffness  $\geq 2.90 \text{ kPa}$
- Platelet count  $\geq 150,000/\text{mm}^3$ ;
- Albumin  $\geq 3.3$  g/dL;
- Creatinine Clearance (CL<sub>cr</sub>) as calculated by the Cockcroft-Gault equation  $\geq$  90 ml/min;

### **Exclusion Criteria:**

- Pregnant or lactating females;
- ALT > 5X ULN;
- Other causes of liver disease including autoimmune, viral, and alcoholic liver disease;
- Cirrhosis of the liver as defined by any of the following:
  - a. Cirrhosis on historical liver biopsy (eg, Brunt/Kleiner stage 4 or equivalent)
  - b. Evidence of cirrhosis on liver imaging (eg, ultrasound, CT, or MRI) including a nodular liver surface, splenomegaly, or portal venous collaterals
  - c. Screening FibroSURE/FibroTest  $^{\circledR} \ge 0.75$ , as determined by the central laboratory
  - d. Prior history of decompensated liver disease, including ascites, hepatic encephalopathy, or variceal bleeding;
- BMI  $< 18 \text{ kg/m}^2$ ;
- Uncontrolled diabetes mellitus (hemoglobin A1c > 9% at screening);
- INR > 1.2 unless on anticoagulant therapy;
- Total bilirubin > 1x ULN, except with diagnosis of Gilbert's syndrome.

Refer to Sections 4.2 and 4.3 for complete listing of inclusion and exclusion criteria.

# Study Procedures/ Frequency:

After signing the informed consent form, subjects will complete a screening visit which will include the following assessments: complete medical history, physical examination (PE), vital signs, laboratory assessments (blood chemistry, hematology, coagulation panel, hemoglobin A1c, biomarkers), viral serology, pregnancy test (for females of child-bearing potential), standard 12-lead ECG, MRI-PDFF and MRE examinations, urine drug test, review of concomitant medications and adverse events.

After the screening period and a randomization visit at Baseline/Day 1, study visits will occur on Weeks 1, 4, 8, 12, 16, 20 and 24 with a Follow-Up visit 4 weeks after the last dose of study drug. At minimum, vital signs, symptom driven PE, safety laboratory tests (blood chemistry, hematology, and coagulation panel), review of concomitant medications and adverse events will be done at every visit.

Eligible subjects will be randomized to one of 3 treatment groups. Prior to initial dosing, required Baseline/Day 1 assessments will be performed

and will include Quality of Life (QoL) assessments (general and pruritus), symptom driven PE, vital signs, laboratory assessments, pregnancy tests (for females of child-bearing potential), urine, blood, and stool collection for biomarker assessment, single PD sampling, standard 12-lead ECG, FibroScan®, review of concomitant medications and adverse events

#### PPD

Subjects will return to clinic for a safety visit at Week 1. Week 1 assessments include QoL: pruritus assessments, symptom driven PE, vital signs, and laboratory tests (blood chemistry, hematology, coagulation panel, lipid profile, biomarkers, PK and PD sampling).

While on study, subjects will undergo the following procedures and laboratory assessments:

- MRE and MRI-PDFF at Weeks 12 and 24
- FibroScan<sup>®</sup> at Baseline/Day 1 and Weeks 12 and 24
- Single PK and PD sampling at Baseline/Day 1 (PD only) and at Weeks 1, 4, 8, 12, 16, 20, and 24
- Blood for Biomarkers at Baseline/Day 1, and Weeks 1, 4, 12, and 24
- 12-lead ECGs at Baseline/Day 1, and Weeks 12 and 24
- Blood chemistry, hematology, coagulation panel, and fasting lipid profile at Baseline/Day 1 and at Weeks 1, 4, 8, 12, 16, 20, and 24
- Hemoglobin A1c (HbA1c) at Baseline/Day 1, Weeks 12 and 24
- Stool collection at Baseline/Day 1 and Week 24
- Urine collection at Baseline/Day 1 and Weeks 1, 4, 12, and 24
- Urine pregnancy test (females of childbearing potential only) at Baseline/Day 1 and Weeks 4, 8, 12, 16, 20, and 24
- QoL: general assessments [SF-36 health survey, Chronic Liver Disease Questionnaire (CLDQ), and Work Productivity and Activity Impairment (WPAI)] at Baseline/Day 1 and Weeks 12 and 24
- QoL: pruritus assessments (VAS-itch and 5D-itch) at Baseline/Day 1 and Weeks 1, 4, 8, 12, 16, 20, and 24

Subjects will return for their final visit, the Follow-Up visit, 4 Weeks after the last dose of study drug. At this visit assessments include a symptom driven PE, vital signs, safety laboratory tests, and review of concomitant medications and adverse events. A urine pregnancy test will be performed for females of child bearing potential only.

| | PPD |
|---|---|
| Test Product: | GS-9674 30 mg tablet administered orally once daily with food. |
| | GS-9674 100 mg tablet administered orally once daily with food. |
| Reference Product: | Placebo-to-match (PTM) GS-9674 30 mg tablet administered orally once daily with food. |
| | Placebo-to-match (PTM) GS-9674 100 mg tablet administered orally once daily with food. |
| Dose and Mode of Administration: | • Treatment Group A: GS-9674 30 mg (1 x 30 mg tablet) + PTM GS-9674 100 mg (1 x PTM 100 mg tablet) administered orally once daily with food |
| | <ul> <li>Treatment Group B: GS-9674 100 mg (1 x 100 mg tablet) + PTM GS-9674 30 mg (1 x PTM 30 mg tablet) administered orally once daily with food</li> </ul> |
| | • Treatment Group C: PTM GS-9674 30 mg (1 x PTM 30 mg tablet) + PTM GS-9674 100 mg (1 x PTM 100 mg tablet) administered orally once daily with food |

## Criteria for Evaluation:

Safety:

The primary endpoint is the safety of GS-9674 in subjects with NASH. Safety will be assessed during the study through the reporting of AEs,

and by clinical laboratory tests and vital sign assessments at various time points during the study. Concomitant medication usage will also be assessed throughout the study.

An independent, external Data Monitoring Committee (DMC) that consists of two hepatologists and a PhD statistician will convene once 20 subjects have been enrolled and every 3 to 4 months thereafter to monitor the study for safety events. The DMC will meet on an ad hoc basis if there are at least 3 Grade ≥ 3 serious, treatment-related Common Terminology Criteria for Adverse Events (CTCAE) observed in the study. In the event of two similar Grade 4-CTCAE treatment-related adverse events or one Grade 5-CTCAE treatment-related adverse event, the DMC will review the data and advise the sponsor regarding stopping or continuing the study.

| Efficacy: | Efficacy will be assessed through a number of exploratory endpoints. These exploratory endpoints are described in Section 8.1.3. |
|---|---|
| Pharmacokinetic and<br>Pharmacodynamic: | Plasma concentrations of GS-9674, GS-716070 (metabolite of GS-9674), and other metabolites as appropriate, will be determined for PK analyses as applicable. Plasma or serum concentrations of FGF19, C14, and bile acids will be determined as applicable for PD analyses. |
| Statistical Methods: | |
| Safety Analysis: | All safety data collected will be listed and summarized, as appropriate, by treatment group. |
| Efficacy<br>Analysis: | The biological activity of GS-9674 will be evaluated using biomarker variables. PPD |
| Exploratory<br>Analysis: | PPD |
| Sample Size: | Due to the exploratory nature of this study, no formal power calculations were used to determine sample size. The number of subjects was chosen based on clinical experience with other similar proof of concept studies. |

This study will be conducted in accordance with the guidelines of Good Clinical Practice (GCP) including archiving of essential documents.

## GLOSSARY OF ABBREVIATIONS AND DEFINITION OF TERMS

Ab antibody
AE adverse event

ALP alkaline phosphatase
ALT alanine aminotransferase

Apo B apolipoprotein B

aPTT activated partial thromboplastine time

AST aspartate aminotransferase ATP adenosine triphosphate

ATV atorvastatin

AUC area under the plasma/serum concentration versus time curve

AUC<sub>tau</sub> area under the plasma/serum concentration versus time curve over the dosing

interval

AUC<sub>inf</sub> area under the plasma/serum concentration versus time curve extrapolated to

infinite time, calculated as AUC<sub>0-last</sub> + ( $C_{last}/\lambda_z$ )

AUC<sub>partial</sub> partial area under the plasma/serum concentration versus time curve

BAP Biomarker Analysis Plan

BCRP breast cancer resistance protein

BMI body mass index
BUN blood urea nitrogen

BW body weight

C4 7-alpha-hydroxy-4-cholesten-3-one

CBC complete blood count cc cubic centimeter

CFR code of federal regulations

CI confidence interval
CK-18 cytokeratin 18
CL systemic clearance
CL<sub>cr</sub> creatinine clearance

CLDQ Chronic Liver Disease Questionnaire

C<sub>last</sub> last observed quantifiable plasma/serum concentration of the drug

 $C_{max}$  maximum observed plasma/serum concentration of drug  $C_{min}$  minimum observed plasma/serum concentration of drug  $C_{tau}$  observed drug concentration at the end of the dosing interval

CRO contract (or clinical) research organization

CsA cyclosporine

CSR Clinical Study Report

CTCAE Common Terminology Criteria for Adverse Events

CV cardiovascular CYP cytochrome P450 Gilead Sciences, Inc.

Final Amendment 1

CYP2C8 cytochrome P4502C8
CYP3A cytochrome P4503A

DAB metabolite of dabigatran etexilate

DDI drug-drug interaction

DE dabigatran etexilate

DILI drug induced liver injury

DMC Data Monitoring Committee

DNA deoxyribonucleic acid

DSPH Drug Safety and Public Health

EC ethics committee

EC<sub>50</sub> concentration of drug that gives half-maximal response

ECG electrocardiogram

eCRF electronic case report form EDC electronic data capture  $ELF^{TM}$  Test enhanced liver fibrosis test

ET early termination
EU European Union

ESA erythropoiesis-stimulating agent

FAS Full Analysis Set

FDA (United States) Food and Drug Administration

FGF19 fibroblast growth factor 19 FSH follicle-stimulating hormone

FXR farnesoid X receptor GCP good clinical practice

GCSF granulocyte colony stimulating factor

GFZ gemfibrozil

GGT gamma glutamyl transferase

GSI Gilead Sciences, Inc.

Hb hemoglobin HbA1c hemoglobin A1c

HBsAg hepatitis B surface antigen

HBV hepatitis B virus

HCC hepatocellular carcinoma hCG human chorionic gonadotropin

HCV hematocrit hepatitis c virus

HDPE high-density polyethylene
HIV human immunodeficiency virus
HIV-1 human immunodeficiency virus type 1

HLT high-level term

Protocol GS-US-402-1852 Final Gilead Sciences, Inc. Amendment 1

HLGT high-level group term

HMG-CoA 3-hydroxy-3-methylglutaryl-coenzyme A
HOMA-IR homeostatic assessment of insulin resistance

IB investigator's brochure ICF informed consent form

ICH International Conference on Harmonization of Technical Requirements for

Registration of Pharmaceuticals for Human Use

ID identification

IEC independent ethics committee/ institutional ethics committee

IND Investigational New Drug (Application)

INR international normalized ratio
IRB institutional review board

IUD intrauterine device

IWRS interactive web response system

LDH lactate dehydrogenase LLT lower-level term

MedDRA Medical Dictionary for Regulatory Activities

MCV mean corpuscular volume

MDZ midazolam

miRNA micro ribonucleic acid mm Hg millimeters of mercury

MRE magnetic resonance elastography
MRI magnetic resonance imaging

MRI-PDFF magnetic resonance imaging – proton density fat fraction

NAFLD nonalcoholic fatty liver disease

NAS NAFLD Activity Score
NASH nonalcoholic steatohepatitis

NMR nuclear magnetic resonance spectroscopy

NOAEL no observed adverse event level

OATP organic anion-transporting polypeptide

oz ounce

PBC primary biliary cholangitis

PD pharmacodynamic
PE physical exam
PK pharmacokinetic
P-gp P-glycoprotein
pH measure of acidity

PRA pravastatin

PSC primary sclerosing cholangitis

PT preferred term

Final Amendment 1

PT prothrombin time PTM placebo-to-match

PTT partial prothrombin time

QA quality assurance
QD once a day
QoL quality of life
RBC red blood cell count

RIF rifampin

RNA ribonucleic acid

ROS reactive oxygen species, or

rosuvastatin

SADR serious adverse drug reaction

SAE serious adverse event
SAP statistical analysis plan
SD standard deviation

SF-36 Short Form (36) Health Survey

SOC system organ class

SOP standard operating procedure

SUSAR Suspected Unexpected Serious Adverse Reaction

 $t_{1/2}$  An estimate of the terminal elimination half-life of the drug in

serum/plasma/PBMC, calculated by dividing the natural log of 2 by the

terminal elimination rate constant  $(\lambda_z)$ 

TEAE treatment-emergent adverse event  $T_{last} \hspace{1cm} last \hspace{1cm} measured \hspace{1cm} concentration \\ T_{max} \hspace{1cm} time \hspace{1cm} (observed \hspace{1cm} time \hspace{1cm} point) \hspace{1cm} of \hspace{1cm} C_{max}$ 

TGR5 bile acid receptor TPO thrombopoietin

TR-FRET time-resolved fluorescence resonance energy transfer UGT1A1 uridine diphosphate glucuronosyltransferase 1A1

ULN upper limit of the normal range

US United States

 $\begin{array}{ccc} USPI & & United States product insert \\ V_{ss} & & volume of distribution \\ VAS & & visual analog scale \\ VORI & & voriconazole \\ \end{array}$ 

WBC white blood cell count

WPAI work productivity and activity impairment questionnaire

### 1. INTRODUCTION

## 1.1. Background

Chronic liver disease and the consequences of end-stage liver disease are increasing globally despite improved prevention and treatment of viral hepatitis. This is due to the emerging epidemics of obesity, metabolic syndrome, and diabetes mellitus that are leading to an increased incidence of nonalcoholic fatty liver disease (NAFLD). Nonalcoholic fatty liver disease is characterized by the excess accumulation of lipid droplets within the liver, also known as hepatic steatosis. Prevalence rates of NAFLD range from 6% to 37% worldwide {Vernon et al 2011}, (Ong et al 2007). Nonalcoholic steatohepatitis (NASH), an aggressive form of NAFLD characterized by the presence of inflammation and hepatocellular ballooning, with or without fibrosis, is present in approximately 25% of patients with NAFLD. Nonalcoholic steatohepatitis is associated with increased liver-related mortality (Williams et al 2011), (Ong et al 2007). In the United States (US), it has been estimated that 3% to 6% of the population {Vernon et al 2011}, {Wanless et al 1990}, or the equivalent of up to 15 million adults, have NASH. NASH represents a significant and growing unmet medical need for which there are no currently approved therapies. Furthermore, as NASH is a manifestation of the metabolic syndrome, risk factors for cardiovascular disease (eg. atherosclerotic disease, cardiac arrhythmogenicity) frequently coexist in these patients {Faramawi et al 2008}, {Voulgari et al 2010}, {Dietrich et al 2014}. A treatment that targets the underlying metabolic disorder could potentially ameliorate these cardiovascular risks and associated morbidity and mortality.

Nonalcoholic steatohepatitis is primarily thought to occur as the result of the metabolic syndrome, the impact of obesity, insulin resistance, and dyslipidemia in the liver. Simple steatosis is not sufficient to cause liver injury; it is the presence of inflammation and hepatocellular injury on the background of steatosis that defines NASH and results in the progression to end-stage liver disease and its complications. The "2-hit" hypothesis of NASH suggests that in the setting of steatosis and metabolic dysfunction, increased oxidative stress and the generation of reactive oxygen species (ROS) likely mediate the inflammatory changes in the liver (steatohepatitis) that may lead to progressive fibrosis {Dowman et al 2010}, {Kannel et al 1982}, {Koek et al 2011}, {Sumida et al 2013}. The major pathways in NASH disease progression include those involved in metabolic dysfunction in the hepatocyte, and activation of hepatic stellate cells and macrophages leading to progressive inflammation and liver fibrosis. Advanced fibrosis and cirrhosis are characterized by extensive collagen deposition and remodeling of the extracellular matrix. In addition, evidence suggests that lipotoxic intermediates of fatty acids likely contribute to the etiology of NASH {Neuschwander-Tetri 2010}.

Over time, NASH may result in progressive liver fibrosis, ultimately leading to cirrhosis in 10-20% of affected patients. Advanced fibrosis (bridging fibrosis or cirrhosis) is associated with increased morbidity and mortality {Ekstedt et al 2014}, {Yeh et al 2014}. Patients with cirrhosis may develop hepatocellular carcinoma (HCC) and other complications of end-stage liver disease, including jaundice, fluid retention (edema and ascites), portal hypertension and variceal bleeding, impaired coagulation and hepatic encephalopathy. Decompensated liver disease, as

defined by the development of one of the above complications, has a high mortality and the only known effective treatment is liver transplantation. With the increasing prevalence of obesity and obesity-related diseases, NASH is expected to become the leading indication for liver transplantation, and the leading etiology of HCC among liver transplant recipients in the US {Wong et al 2014}, {Afzali et al 2012}.

### 1.1.1. GS-9674 General Information

GS-9674 is a potent agonist of Farnesoid X Receptor (FXR) whose activity in intestinal epithelial cells results in the release of fibroblast growth factor 19 (FGF19). FGF19 is an endocrine peptide which drives a signaling cascade to decrease lipogenesis, gluconeogenesis, hepatic triglyceride accumulation, and bile acid synthesis. Please refer to the Investigator's Brochure (IB) for additional information on GS-9674, including:

- In vitro FXR agonism
- Nonclinical pharmacokinetics and in vitro metabolism
- Nonclinical pharmacology and toxicology

## 1.1.2. Nonclinical Toxicology

The nonclinical toxicity profile of GS-9674 has been assessed in mice and cynomolgus monkeys administered GS-9674 orally for up to 26 and 13 weeks, respectively. GS-9674-related effects were primarily limited to non-adverse findings in the liver for both species that are likely related to the pharmacology of the compound. Mild increases in alkaline phosphatase (ALP) activity and liver weights were observed in the 4 week and chronic (26 or 13 weeks) studies. In the 4-week studies and 26-week mouse study, these findings were associated with hepatocellular hypertrophy (both species) and minimal oval cell hyperplasia (monkeys). In the chronic monkey study, there were no correlating histological changes in the liver after 13 weeks of dosing. The above findings were observed at  $\geq 100$  mg/kg/day after 4 weeks of dosing and at all doses (> 20 mg/kg/day) after 26 weeks of dosing in mice. In monkeys, the above findings were observed at doses of 300 mg/kg/day after both 4 and 13 weeks of dosing. The decreases in cholesterol (≥ 60 mg/kg/day) and triglycerides (≥ 100 mg/kg/day) as well as increased albumin (≥ 60 mg/kg/day) observed in mice after 4 and/or 26 weeks of dosing as well as the decrease in serum bile acids (300 mg/kg/day) in monkeys after 13 weeks of dosing are also likely to be related to the pharmacology of GS-9674. Other minimal to mild, non-adverse findings observed after 13 or 26 weeks of dosing in monkeys or mice, respectively, that were considered GS-9674related included decreased red blood cell parameters (mouse;  $\geq 20 \text{ mg/kg/day}$ ), increased platelets (mouse; 600/300 mg/kg/day), shortened activated partial thromboplastin time (monkey; 300 mg/kg/day), and increased phosphorus (mouse; 600/300 mg/kg/day). All findings observed in monkeys after 13 weeks of dosing had resolved at the end of the 4-week recovery period. The no-observed-adverse effect levels (NOAEL) in mice after 26 weeks of dosing and in monkeys after 13 weeks of dosing were 60 and 300 mg/kg/day, respectively.

Preliminary PK data from Cohort 5 (administration of GS-9674 100 mg with food) in the ongoing Phase 1 study of GS-9674 (GS-US-402-1851, included in IB, Ed 02) indicate adequate safety margins based on GS-9674 exposures at the nonclinical NOAEL doses in mouse and cynomolgus monkey (Table 1-1).

Table 1-1. Exposure Margins for GS-9674 Based on Observed GS-9674 Exposure After Administration of 100 mg GS-9674 Under Fed Conditions in Cohort 5 Compared to Exposures Observed at NOAEL Doses in Mouse and Cynomolgus Monkey

| | NO | | |
|---|---|---|---|
| Species | Dose<br>mg/kg/day | AUC <sub>tau</sub><br>μg*hr/mL | Exposure Margin <sup>a</sup> |
| Mouse | 60 | Male: 66<br>Female: 110 | Male: 13<br>Female: 22 |
| Cynomolgus Monkey | 300 | 110 | 22 |

a Calculated using observed human AUC $_{inf}$  of 5.02  $\mu g*hr/mL$  at 100 mg QD dose administered fed from Cohort 5 in Study GS-US-402-1851.

# 1.1.3. Nonclinical Pharmacology

GS-9674 is a potent and selective agonist of FXR. This conclusion is supported by the following data: 1) modeling demonstrated an interaction of GS-9674 with the binding domain of FXR consistent with agonist activity, 2) GS-9674 induced an agonist response in a time-resolved fluorescence resonance energy transfer (TR-FRET) biochemical assay with an EC<sub>50</sub> of 16 nM, which was comparable to that of other known FXR agonists, and 3) GS-9674 did not activate the structurally similar bile acid receptor TGR5, did not activate other nuclear hormone receptors, and did not bind to a panel of other off-target receptors and enzymes.

The cellular potency of GS-9674 to activate FXR-mediated transcription was characterized using a firefly luciferase reporter gene engineered under the control of a FXR/RXR response element (PC-402-2012). GS-9674 caused complete FXR activation with an EC<sub>50</sub> value of 43 nM, which was more potent than chenodeoxycholic acid (EC<sub>50</sub> of 1770 nM).

Oral dose-ranging experiments in male cynomolgus monkeys demonstrated maximal increases in plasma FGF19 at a dose of 5 mg/kg (PC-402-2016). In addition, the oral administration of GS-9674 (30 mg/kg) to cynomolgus monkeys directly activated intestinal FXR, as measured by the expression of FXR-target genes in the ileum (15-fold increase in FGF19 mRNA, and a 2-fold increase in organic solute transporter (OST) $\alpha$  and (OST) $\beta$  mRNA) (PC-402-2005).

The effects of GS-9674 on FGF19 levels were compared in cynomolgus monkeys following both oral and intravenous (IV) administration (PC-402-2016). Despite greater exposures following IV administration, only the oral administration of GS-9674 increased circulating FGF19 levels. These data suggest that intestinal FXR agonism by GS-9674 causes FGF19 production, whereas low systemic free drug concentrations limit effects following IV administration of GS-9674.

GS-9674 was evaluated in a choline-deficient high fat diet /NaNO<sub>2</sub> rat model of liver fibrosis (PC-402-2015). This in vivo model utilized "2 hits" to mimic the metabolic and oxidative stress components of NASH disease in humans {Nakamoto et al 2009}, {Murakami et al 2013}. Treatment with GS-9674 dose-dependently reduced both biochemical and histological measures of liver fibrosis in this model.

Safety pharmacology studies have been conducted to examine the potential effects of GS-9674 on the cardiovascular (CV), respiratory, and central nervous system (CNS) systems. There were no GS-9674-related effects on the CNS or respiratory system in mice administered up to 600 mg/kg. In addition, there was no significant human ether-a-go-go-related gene inhibition at concentrations up to  $100~\mu M$  or GS-9674-related effects on the CV system in monkeys administered up to 300~mg/kg.

Overall, the results from these pharmacology studies demonstrate that GS-9674 is a potent and selective agonist of intestinal FXR with the potential to benefit NASH patients by inducing FGF19 production.

#### 1.1.4. Nonclinical Pharmacokinetics

GS-9674 has shown low oral bioavailability in nonclinical species (approximately 10% and 20% when dosed as PPD ). Low, pH-dependent solubility and efflux transport have been identified as factors likely limiting GS-9674 absorption.

The low systemic clearance (CL) of GS-9674 in rats, dogs and monkeys was considerably lower than the predicted hepatic clearance based on in vitro studies with hepatocytes. This discrepancy is most likely a result of protein-restricted clearance in vivo due to the very high plasma protein binding (> 99.6%) across species. The volume of distribution ( $V_{ss}$ ) of GS-9674 was consistent with extracellular fluid (ranging from 0.16-0.21 L/kg) in rats, dogs, and monkeys.

After oral dosing to albino and pigmented mice, [<sup>14</sup>C]GS-9674-derived radioactivity was distributed to most of the tissues, with the highest maximum concentrations of radioactivity determined in organs of absorption and excretion. Generally similar distribution patterns and tissue concentrations of [<sup>14</sup>C]GS-9674-derived radioactivity were observed in albino and pigmented mice with no observed binding to melanin. In both strains, no quantifiable radioactivity was detected in brain, suggesting [<sup>14</sup>C]GS-9674-derived radioactivity did not cross the blood:brain barrier. Fecal elimination was a predominant route of elimination of [<sup>14</sup>C]GS-9674-derived radioactivity in both mice (85.7% and 5.45% recovered in feces and urine, respectively) and monkeys (78.2% and 69.7% recovered in feces in intact and bile duct cannulated animals) likely representing drug not absorbed from the gastrointestinal tract. Approximately 6% of the administered radioactivity was excreted in bile and urine in monkeys. Radiolabeled material was primarily excreted within the first 48 hours.

GS-9674 undergoes oxidative metabolism in human hepatocytes. Comparison of metabolism in hepatocytes from mice, rats, dogs, monkeys, and humans did not identify any metabolites unique to humans, supporting the selection of mice and monkeys for the assessment of the toxicology of GS-9674. Of the recombinant human CYP isozymes tested, CYP2C8, CYP3A4, and CYP2C19 were shown to metabolize GS-9674. Potent inhibitors of these CYPs therefore may affect metabolism of GS-9674. GS-9674 had little inhibitory effect on the activities of CYP1A2, CYP2B6, CYP2C19 or CYP2D6 (IC<sub>50</sub> > 25  $\mu$ M). For CYP2C8, CYP2C9, and CYP3A, IC<sub>50</sub> values of 2.4 to 13.6 µM were obtained but GS-9674 was not a mechanism-based inhibitor of these enzymes, GS-9674 showed moderate inhibition of human UGT1A1, sodium-taurocholate cotransporting polypeptide (NTCP), and bile salt export pump (IC<sub>50</sub> 2.8-7.7 µM). GS-9674 inhibited human OATP1B1, OATP1B3, and OATP2B1 with IC<sub>50</sub> values of 0.68, 0.41, and 0.21 µM, respectively. GS-9674 therefore has the potential to affect hepatic/intestinal uptake of OATP substrates or metabolism of CYP2C8, CYP2C9, or CYP3A4 substrates when its concentrations are sufficiently high. However, low solubility, high protein binding (> 99.98%) and low systemic levels reduce the potential for GS-9674 to cause drug-drug interactions via inhibition of metabolic enzymes and transporters.

GS-9674 is a substrate for efflux transporters P-glycoprotein and breast cancer resistance protein, as well as the uptake transporters OATP1B1, 1B3, and 2B1, and NTCP. Inhibitors or genetic polymorphisms affecting the activity of these transporters may affect GS-9674 intestinal absorption and hepatic uptake. This was illustrated in an in vivo study in monkeys where pretreatment with cyclosporin A, a known inhibitor of efflux transporters, increased the bioavailability of GS-9674 approximately 5-fold.

GS-9674 is highly selective for FXR over other nuclear hormone receptors in cell-based reporter assays, including those associated with potential for induction of human drug metabolizing enzymes and transporters (eg, pregnane X receptor, constitutive androstane receptor). Thus the liability of GS-9674 to cause drug-drug interactions through proteins regulated by these nuclear receptors is low.

#### 1.1.5. Clinical Trials of GS-9674

As of 23 September 2016, 4 Phase 1 clinical studies are ongoing (GS-US-402-1851, GS-US-402-3885, GS-US-402-2102, and GS-US-402-2101), and 4 Phase 2 studies in subjects with NAFLD, NASH, PBC, and PSC are ongoing or planned (GS-US-384-3914, GS-US-402-1852, GS-US-427-4024, and GS-US-428-4025, respectively). These Phase 1 and 2 studies are described in the IB.

A brief summary of preliminary results not included in the IB from ongoing study GS-US-402-2102 is presented below.

### 1.1.5.1. GS-US-402-2102

Study GS-US-402-2102 is an ongoing Phase 1, open-label, multicenter, multiple-cohort study designed to evaluate transporter and CYP-mediated drug-drug interactions (DDIs) between GS-9674 100 mg and various probe drugs in healthy subjects. A total of approximately 180 subjects are planned to be enrolled.

Preliminary PK results from the following cohorts are presented below and in Table 1-2 and Table 1-3:

- Cohort 1: Impact of OATP/MRP2/P-gp inhibition (single dose cyclosporine 600 mg: CsA) or OATP1B1/1B3 inhibition (single dose rifampin 600 mg: RIF) on single dose administration of GS-9674 100 mg with food (N=24). Single doses of CsA or RIF significantly increased GS-9674 exposure (6.5- and 8.0-fold respectively), with more modest increases in GS-716070 exposure (3.3- and 4.9-fold respectively). These data indicate the GS-9674 is a sensitive substrate of hepatic OATP with intestinal P-gp playing a minimal to no role in GS-9674 absorption as seen by a smaller increase in GS-9674 by CsA compared to single dose RIF. Based on these data, coadministration of GS-9674 with potent inhibitors of OATP is not recommended and moderate inhibitors of OATP should be used with caution, whereas GS-9674 may be coadministered with P-gp inhibitors.
- Cohort 2: Impact of CYP3A inhibition (multiple dose voriconazole 200 mg BID 4 days: VORI) and CYP2C8 inhibition (multiple dose gemfibrozil 600 mg BID 4 days: GFZ) on single dose administration of GS-9674 100 mg with food (N=18). Coadministration of GS-9674 with VORI did not result in clinically meaningful changes in GS-9674 or GS-716070 exposures indicating that CYP3A plays a minimal role in the disposition of GS-9674 and GS-716070. As such, GS-9674 may be coadministered with CYP3A inhibitors. Coadministration of GS-9674 with GFZ increased GS-9674 exposure 75% with reduction of GS-716070 exposure by 55% indicating that biotransformation of GS-9674 to GS-716070 is predominantly mediated by CYP2C8. Based on the less than 2-fold increase in GS-9674 exposure, GS-9674 may be coadministered with inhibitors of CYP2C8.
- Cohort 3: Impact of CYP3A/2C8/OATP/P-gp induction (multiple dose rifampin 600 mg QD 7 days in the evening: RIF) on single dose AM administration of GS-9674 100 mg with food (N=18). Plasma exposure of GS-9674 and GS-716070 were substantially reduced after multiple dose administration of RIF indicating that GS-9674 and GS-716070 are sensitive to induction of OATP and CYP2C8. As such, coadministration of GS-9674 with potent or moderate inducers of OATP or CYP2C8 is not recommended.
- Cohort 5: Impact of single dose administration of GS-9674 100 mg with food on CYP3A activity (single dose midazolam: MDZ) or OATP/CYP3A activity (single dose atorvastatin: ATV) (N=24). GS-9674 did not alter MDZ exposure (90%CIs of the %GMR for AUC and C<sub>max</sub> were contained within the predetermined lack of effect bounds of 70-143%) indicating the GS-9674 is not an inhibitor of CYP3A. As such, GS-9674 may be coadministered with CYP3A substrates. GS-9674 modestly increased ATV exposure (39%). Similar increases in

ATV exposure do not necessitate a priori dose modification as per the LIPITOR® United States product insert (USPI). As such, ATV may be coadministered with GS-9674

• Cohort 6: Impact of single dose administration of GS-9674 100 mg with food on P-gp (single dose dabigatran etexilate 75 mg: DE), OATP (single dose pravastatin 40 mg: PRA) or OATP/BCRP (single dose rosuvastatin 10 mg: ROS) (N=24). GS-9674 did not alter DE (free or total dabigatran: DAB metabolite of DE), PRA, or ROS exposures (90%CIs of the %GMR for AUC and C<sub>max</sub> were contained within the predetermined lack of effect bounds of 70-143%) indicating the GS-9674 is not an inhibitor of P-gp, OATP, or BCRP. As such, GS-9674 may be coadministered with P-gp, OATP, or BCRP substrates.

Table 1-2. Preliminary Pharmacokinetic Results from Study GS-US-402-2102 Evaluating the Effect of DDIs on Administration of 100 mg GS-9674 with Food (Cohorts 1-3)

| | | %GMR (90%CI) Test/Reference | | | | |
|---|---|---|---|---|---|---|
| | | Cohort | 1 (N=24) | Cohort | 2 (N=18) | Cohort 3 (N=18) |
| Analyte | PK<br>Parameter | CsA | RIF <sup>a</sup> | VORI | GFZ | RIFb |
| CS 0(74 | $AUC_{inf}$ | 655<br>(577, 743) | 796<br>(719, 880) | 95.9<br>(81.0, 114) | 175<br>(149, 206) | 32.8<br>(27.9, 38.4) |
| GS-9674 | $C_{max}$ | 512<br>(448, 584) | 547<br>(497, 603) | 76.8<br>(60.2, 97.9) | 139<br>(115, 168) | 35.5<br>(29.1, 43.3) |
| CS 71(070 | AUC <sub>inf</sub> | 331<br>(297, 369) | 493<br>(442, 551) | 129<br>(109, 154) | 44.5<br>(38.7, 51.1) | 12.6<br>(10.5, 15.0) |
| GS-716070 | $C_{max}$ | 211<br>(191, 232) | 301<br>(274, 331) | 99.2<br>(81.1, 121) | 31.2<br>(26.1, 37.4) | 17.0<br>(13.7, 21.2) |

Data are presented to 3 significant digits

a Single Dose

b Multiple Dose

Table 1-3. Preliminary Pharmacokinetic Results from Study GS-US-402-2102 Evaluating the Effect of GS-9674 100 mg with Food on CYP3A, OATP/CYP3A, P-gp, OATP, or OATP/BCRP (Cohorts 5-6)

| Cohort | Enzyme/<br>Transporter | Analyte | PK Parameter | Test | Reference | % GMR<br>(90%CI)<br>Test/Reference |
|---|---|---|---|---|---|---|
| | CATEDA | 1.00 | $AUC_{inf}$ | 37.3 (27.5) | 63.9 (29.1) | 102 (95.8, 108) |
| 5 | CYP3A | MDZ | $C_{max}$ | 7.79 (27.6) | 7.92 (35.6) | 100 (94.8, 106) |
| (N=24) | OATP/ | ATV | $AUC_{inf}$ | 15.5 (33.5) | 10.8 (39.0) | 139 (124, 156) |
| | CYP3A | ATV | $C_{\text{max}}$ | 1.06 (35.6) | 0.98 (35.9) | 107 (94.6, 120) |
| | P-gp | Total<br>DAB | $AUC_{inf}$ | 624 (32.0) | 535 (34.3) | 118 (109, 128) |
| | | | $C_{max}$ | 84.4 (40.0) | 68.0 (37.8) | 125 (112, 139) |
| | | Free<br>DAB | $\mathrm{AUC}_{\mathrm{inf}}$ | 543 (32.0) | 477 (37.3) | 116 (108, 124) |
| 6 | | | $C_{max}$ | 75.0 (39.6) | 60.8 (42.5) | 125 (114, 138) |
| (N=24) | OATP | PRA | $AUC_{inf}$ | 109 (55.6) | 99.6 (66.7) | 115 (104, 126) |
| | | | $C_{max}$ | 41.7 (58.8) | 42.4 (66.5) | 104 (91.5, 117) |
| | OATP/ | ROS | $AUC_{inf}$ | 38.3 (40.3) | 34.9 (39.5) | 111 (101, 121) |
| | BCRP | | $C_{max}$ | 3.06 (40.4) | 2.86 (43.4) | 108 (98.3, 119) |

Data are presented as mean (%CV) to three significant digits

## 1.2. Rationale for This Study

Current evidence suggests that NASH is a consequence of the metabolic syndrome with resulting lipotoxicity and oxidative stress in the steatotic liver, setting off an inflammatory response with subsequent activation of hepatic stellate cells and fibrogenesis. FXR agonism has been shown to reduce hepatic lipid synthesis and circulating triglycerides due to down regulation of SREBP-1c, as well as reduce insulin resistance and hepatic gluconeogenesis. Thus GS-9674 is postulated to halt the instigating triggers for NASH. Animal models have demonstrated the ability for GS-9674 to reverse the metabolic dysfunction and NASH-like liver injury in a choline-deficient high fat diet /NaNO<sub>2</sub> rat model of liver fibrosis. This Phase 2 study has been designed as a multicenter, randomized, double-blind, placebo-controlled study evaluating the safety and efficacy of GS-9674 for 24 weeks in subjects with NASH. Approximately 125 NASH subjects without cirrhosis will be randomized in a 2:2:1 ratio to receive GS-9674 at a dose of 30 mg or 100 mg orally QD, or placebo. Randomization will be stratified by the presence or absence of diabetes mellitus, a common comorbidity in patients with this condition.

Inclusion criteria for the study were developed in order to noninvasively identify subjects with NASH. Specifically, all subjects will have a clinical diagnosis of NAFLD, evidence of  $\geq 10\%$  hepatic steatosis on MRI-PDFF {Bannas et al 2015}, and increased liver stiffness on MRE ( $\geq 2.90$  kPa). Previous studies have shown that patients with NAFLD and increased liver stiffness by MRE have a high probability of NASH on liver biopsy {Loomba et al 2014}, {Chen et

al 2011}. For example, Chen et al. reported that an MRE liver stiffness cut-off of  $\geq$  2.90 kPa was 83% sensitive, 82% specific, and had an area under the receiver operating characteristic curve (AUROC) of 0.93 and positive predictive value of 88% for the differentiation of simple steatosis from NASH on biopsy. Moreover, in a meta-analysis of MRE for the diagnosis of NAFLD-related fibrosis {Singh et al 2016}, a liver stiffness  $\geq$  2.88 kPa optimally identified the presence of at least stage 1 fibrosis (AUROC 0.86). Based on these criteria, subjects enrolled in this study have a high probability of NASH with fibrosis, a population with a large unmet medical need. Since the safety and PK of GS-9674 have not yet been explored in subjects with cirrhosis, criteria have been developed in order to exclude cirrhotic subjects based on a validated serum marker for fibrosis (FibroSURE/FibroTest\*) and historical clinical, histological, and imaging data {Ratziu et al 2006}.

The primary endpoint of this study will be the safety and tolerability of GS-9674. In addition, the biological activity of GS-9674 will be determined based on endpoints including routine liver biochemistry (eg, ALT and GGT); noninvasive serum markers of liver injury (eg, serum CK-18, FibroSURE/FibroTest® and ELF™ Test); and imaging-based methods for quantifying hepatic steatosis (MRI-PDFF) and fibrosis (MRE and FibroScan®). An important endpoint of interest is the proportion of subjects achieving ≥ 30% reduction in steatosis as assessed by MRI-PDFF. This level of reduction has been associated with a significant improvement in NASH histology (≥ 2-point reduction in NAFLD Activity Score) {Patel et al 2015}. Based on preclinical and clinical data, a treatment duration of 24 weeks with GS-9674 is expected to be sufficient to lead to meaningful improvements in hepatic steatosis on MRI-PDFF and liver biochemistry. In addition to these liver-related endpoints, the effects of GS-9674 on carbohydrate and lipid metabolism (eg, glucose, insulin, free fatty acids, apolipoproteins, lipid profiles, and metabolites) will be closely monitored in light of the mechanism of action of GS-9674 and the importance of metabolic dysfunction in contributing to the morbidity and mortality (eg, cardiovascular) of subjects with NASH.

This study will evaluate the safety, tolerability, and efficacy of 30 mg and 100 mg GS-9674 administered with food for 24 weeks in subjects with NASH. The doses were selected based on short-term safety, PK and PD results from Study GS-US-402-1851 in healthy subjects.

Across the range of GS-9674 doses evaluated (10-300 mg QD), doses  $\geq$  30 mg provide comparable intestinal FXR activation assessed as increases in FGF19 exposure. Food, by slowing oral absorption of GS-9674, results in prolonged elevation of plasma FGF19 concentrations. Exposure-response relationships show that changes in C4 exposure are negatively correlated with changes in FGF19 exposure as well as GS-9674 exposure. Based on these results, GS-9674 doses of 30 and 100 mg with food are selected for further study as they are expected to 1) provide enteral FXR agonism and improvements in subjects with NASH and 2) inform on the impact of increasing systemic GS-9674 exposure on safety and efficacy.

In the Phase 1 study, GS-US-402-1851, GS-9674 was tested at doses up to 300 mg once daily for up to 14 days and was well tolerated. Taken together, these data support the evaluation of GS-9674 30 and 100 mg in subjects with NASH.

# 1.3. Risk/Benefit Assessment for the Study

This study will provide information on the safety and efficacy of GS-9674 for the treatment of patients with NASH. As there are currently no approved therapies for NASH, there is a large unmet medical need for this growing population of patients.

Subjects with NASH randomized to the placebo control arm in the study may benefit from frequent medical monitoring and close assessment of their NASH during the duration of placebo treatment. Subjects randomized to GS-9674 may benefit from an improvement in their underlying NASH which may manifest as improvements in liver biochemistry, measures of hepatic steatosis or fibrosis, or improvements in quality of life. Importantly, this study will provide further data to inform the clinical development of the investigational medicinal product GS-9674 for use in an area of unmet medical need.

In the Phase 1 study, 94 subjects have received GS-9674 in single or multiple doses (14 days) up to 300 mg. All treatment emergent adverse events (TEAEs) were mild to moderate (Grade 1 or 2), and overall, the rate of any adverse events (AEs) was similar between subjects treated with GS-9674 or placebo. The predominant toxicities were anemia, back pain, diarrhea, and headache. Grade 2 or 3 elevations in serum ALT were seen in five (5%) GS-9674 treated subjects and one (4%) placebo treated subject. Grade 2 or 3 ALT elevations that occurred on-treatment were observed in 2/23 (9%) BID treated subjects, but none of the 71 subjects who received once daily (QD) GS-9674 dosing. In these cases, elevations in serum bilirubin or prolongation of INR were not observed, serum ALT levels normalized upon treatment cessation, and no evidence of drug hypersensitivity syndrome (eg, fever, rash, eosinophilia) was noted. In nonclinical studies, effects on the liver have been limited to non-adverse mild increases in alkaline phosphatase and liver weights and minimal hepatocellular hypertrophy that are likely a pharmacological response to FXR agonism. There were no elevations in liver transaminases or changes in liver pathology (degeneration/necrosis) in the nonclinical studies to suggest direct cellular damage. In order to mitigate the potential risk of hepatotoxicity with GS-9674, QD dosing of GS-9674 has been chosen for this study. Moreover, close monitoring of liver biochemistry values will be performed and parameters for discontinuation of the study drugs due to liver test abnormalities have been defined (see Section 7.5, Toxicity Management: Observation for Drug-Induced Liver Injury) and will be closely followed.

Additional risks to study subjects include those attributable to study participation in general, including risks associated with frequent clinic visits and laboratory blood draws, and the associated pain and discomfort of phlebotomy. Strategies to mitigate these risks include close monitoring of lab values as well as AEs. Parameters for discontinuation of the study drugs due to AEs and non-hepatic laboratory abnormalities are also defined and will be closely followed.

Overall, the nonclinical and limited preliminary clinical data show a positive benefit/risk ratio in support of the study in subjects with NASH. Appropriate safety monitoring will be conducted throughout the study to further characterize the safety profile of GS-9674 in NASH subjects without cirrhosis.

In summary, there are no approved treatment options available for patients with NASH. Based on past clinical experience with GS-9674, the risk/benefit is positive and supports the continued evaluation of GS-9674 in this patient population. Data from this study will support the development of GS-9674 for the treatment of this condition.

# 1.4. Compliance

This study will be conducted in compliance with this protocol, Good Clinical Practice (GCP), and all applicable regulatory requirements.

# 2. OBJECTIVES

The **primary objective** of this study is as follows:

• To evaluate the safety and tolerability of GS-9674 in subjects with NASH.

The exploratory objectives of this study are as follows:



## 3. STUDY DESIGN

## 3.1. Study Design

This is a Phase 2, randomized, double-blind, placebo-controlled study designed to evaluate the safety, tolerability, and efficacy of GS-9674 in subjects with NASH. To be eligible to participate, subjects must have evidence of hepatic steatosis and increased liver stiffness as assessed by MRI-PDFF and MRE respectively. Any subject with a history of decompensated liver disease, including ascites, hepatic encephalopathy, or variceal bleeding will be ineligible.

The overall study design is presented graphically in Figure 3-1.

Group A (n = 50)GS-9674 30 mg + PTM GS-9674 100 mg Follow Up/End of Study orally once daily **End of Treatment** Randomization Screening Group B (n = 50)GS-9674 100 mg + PTM GS-9674 30 mg orally once daily Group C (n = 25)PTM GS-9674 30 mg + PTM GS-9674 100 mg orally once daily 4 Weeks 4 Weeks 24 Weeks

Figure 3-1. Overall Study Design

PTM = Placebo-to-match

## 3.2. Treatment Plan and Regimen

Subjects meeting the study's entry criteria will be randomly assigned in a 2:2:1 ratio to 1 of 3 different treatment groups (A, B, and C) as shown in Figure 3-1. Randomization will be stratified by the presence or absence of diabetes mellitus as determined by medical history, use of medication for indication of diabetes mellitus, or based on screening lab values if previously undiagnosed (ie, hemoglobin A1c  $\geq$  6.5% OR fasting plasma glucose  $\geq$  126 mg/dL).

Study drug will be administered for a total of 24 weeks from the Baseline/Day 1 visit up to and including the Week 24 visit. Dosage and administration of the study drug and reference product are described in Section 5.3.

## 3.3. Biomarker Testing

## 3.3.1. Biomarker Samples to Address the Study Objectives

Biological specimens will be collected in this study as per the study procedures table

(Appendix 2) PPD

Because biomarker science is a rapidly evolving area of investigation, and adverse events in particular are difficult to predict, it is not possible to specify prospectively all tests that will be done on the specimens provided. The biomarker tests may be modified during or after the end of the study to remove tests no longer indicated and/or to add new tests based upon the growing state of art knowledge. Samples will be

Biomarkers testing can include circulating markers of FXR activity such as FGF19, bile acids, and C4. Circulating protein markers of liver damage and inflammation, lipids, and other biochemicals associated with liver metabolic activity will also be measured. Stool samples may be analyzed for the presence of bile acids and a survey of potential changes in the intestinal microbiome during the study.

### 3.3.2. Biomarker Samples for Optional Future Research

stored for up to 15 years after the end of the study.



# 3.3.3. Biomarker Samples for Optional Genomic Research

PPD



## 4. SUBJECT POPULATION

## 4.1. Number of Subjects and Subject Selection

This study will enroll approximately 125 subjects with nonalcoholic steatohepatitis (NASH).

#### 4.2. Inclusion Criteria

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:

- 1) Males and females between 18-75 years of age; inclusive based on the date of the screening visit;
- 2) Willing and able to give informed consent prior to any study specific procedures being performed;
- 3) Meets all of the following conditions:
  - a. A clinical diagnosis of nonalcoholic fatty liver disease (NAFLD) with histological or imaging evidence of fatty liver within the past two years. If necessary an ultrasound may be performed during screening to confirm NAFLD. Note: criterion a. must be met before evaluating criteria b. and c.
  - b. Screening MRI-PDFF with  $\geq 10\%$  steatosis
  - c. Screening MRE with liver stiffness  $\geq 2.90 \text{ kPa}$ ;
- 4) Platelet count  $\geq 150,000/\text{mm}^3$ ;
- 5) Albumin  $\geq 3.3$  g/dL;
- 6) Creatinine Clearance ( $CL_{cr}$ ) as calculated by the Cockcroft-Gault equation  $\geq 90$  ml/min;
- 7) Female subjects of childbearing potential (see definition in Appendix 4) must have a negative serum pregnancy test prior to starting study treatment;
- 8) All female subjects of childbearing potential who engage in heterosexual intercourse must agree to use a highly effective method of contraception during intercourse from the screening visit throughout the study period and for 30 days following the last dose of study drug (see Appendix 4 for details);
- 9) Female subjects must refrain from egg donation or harvest during treatment and for at least 30 days after last dose of study drug;

- 10) Male subjects are required to use barrier contraception (condom plus spermicide) during heterosexual intercourse from the screening through the study completion and for 90 days following the last dose of study drug (see Appendix 4 for details);
- 11) Male subjects must refrain from sperm donation from screening through at least 90 days following the last dose of study drug;
- 12) Willing and able to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions;
- 13) Must be able to read and complete Quality of Life questionnaires independently.

### 4.3. Exclusion Criteria

Subjects who meet *any* of the following exclusion criteria are not to be enrolled in this study.

- 1) Pregnant or lactating females; lactating females must agree to discontinue nursing before the study drug is administered;
- 2) ALT > 5X ULN;
- 3) Other causes of liver disease including autoimmune, viral, and alcoholic liver disease;
- 4) Cirrhosis of the liver as defined by any of the following:
  - a. Cirrhosis on historical liver biopsy (eg, Brunt/Kleiner stage 4 or equivalent)
  - b. Evidence of cirrhosis on liver imaging (eg, ultrasound, CT, or MRI) including a nodular liver surface, splenomegaly, or portal venous collaterals
  - c. Screening FibroSURE/FibroTest $^{\circ} \ge 0.75$ , as determined by the central laboratory
  - d. Prior history of decompensated liver disease, including ascites, hepatic encephalopathy, or variceal bleeding;
- 5) History of liver transplantation;
- 6) Weight reduction surgery in the past or planned during the study;
- 7) History of intestinal resection or malabsorptive condition that may limit the absorption of GS-9674. Prior cholecystectomy and appendectomy are permitted.
- 8) BMI <  $18 \text{ kg/m}^2$ ;
- 9) Uncontrolled diabetes mellitus (hemoglobin A1c > 9% at screening);
- 10) INR > 1.2 unless on anticoagulant therapy;
- 11) Total bilirubin > 1x ULN, except with diagnosis of Gilbert's syndrome;


- 12) Chronic hepatitis B (HBsAg positive);
- 13) Chronic hepatitis C (HCV RNA positive);
- 14) HIV Ab positive;
- 15) Alcohol consumption greater than 21 oz/week for males or 14 oz/week for females (1oz/30mL of alcohol is present in 1 12oz/360mL beer, 1 4oz/120mL glass of wine, and a 1 oz/30 mL measure of 40% proof alcohol);
- 16) Positive urine screen for amphetamines, cocaine or opiates (ie, heroin, morphine) at screening. Subjects on stable methadone or buprenorphine maintenance treatment for at least 6 months prior to screening may be included in the study. Subjects with a positive urine drug screen due to prescription opioid-based medication are eligible if the prescription and diagnosis are reviewed and approved by the investigator;
- 17) Unstable cardiovascular disease as defined by any of the following:
  - a. Unstable angina within 6 months prior to screening
  - b. Myocardial infarction, coronary artery bypass graft surgery or coronary angioplasty within 6 months prior to screening
  - c. Transient ischemic attack or cerebrovascular accident within 6 months prior to screening
  - d. Obstructive valvular heart disease or hypertrophic cardiomyopathy
  - e. Congestive heart failure;
- 18) History of known hypercoagulable condition or prior arterial or venous thromboembolic disease;
- 19) Use of any prohibited concomitant medications as described in Section 5.5;
- 20) History of a malignancy within 5 years of screening with the following exceptions:
  - a. Adequately treated carcinoma in situ of the cervix
  - b. Adequately treated basal or squamous cell cancer or other localized non-melanoma skin cancer;
- 21) Any laboratory abnormality or condition that could, in the opinion of the investigator, adversely affect the safety of the subject or impair the assessment of study results;

- 22) Participation in another investigational study of a drug or device within 1 month prior or within 5 half-lives of the prior investigational agent (whichever is longer) prior to screening;
- 23) Concurrent participation in another therapeutic clinical study;
- 24) Known hypersensitivity to GS-9674, the metabolites, or formulation excipient;
- 25) Presence of any condition that could, in the opinion of the investigator, compromise the subject's ability to participate in the study, such as history of substance abuse or a psychiatric (including any subjects with a psychiatric hospital admission or emergency room visit in the 2 years prior to screening) or medical condition;
- 26) Unavailable for follow-up assessment or concern for subject's compliance with the protocol procedures;
- 27) Contraindications or inability to complete MRI scanning (eg, presence of permanent pacemakers, implanted cardiac devices, weight restrictions, etc.).

### 5. INVESTIGATIONAL MEDICINAL PRODUCTS

## 5.1. Randomization, Blinding and Treatment Codes

An Interactive Web Response System (IWRS) will be used for centralized randomization and treatment assignment. Randomization will be stratified by the presence or absence of diabetes mellitus as determined by medical history, use of medication for indication of diabetes mellitus, or based on screening lab values if previously undiagnosed (ie, hemoglobin  $A1c \ge 6.5\%$  OR fasting plasma glucose  $\ge 126$  mg/dL).

Investigative site personnel will obtain the subject's identification number and study drug assignment from the IWRS. Subjects and all personnel directly involved in the conduct of the study will be blinded to treatment assignment.

Study drug will be dispensed by the study pharmacist, or designee, in a blinded fashion to the subjects.

## **5.1.1.** Procedures for Breaking Treatment Codes

In the event of a medical emergency where breaking the blind is required to provide medical care to the subject, the investigator (or designee) may obtain treatment assignment directly from the IWRS system for that subject (refer to the Study Reference Binder for IWRS unblinding instructions). Gilead recommends but does not require that the investigator contact the Gilead Medical Monitor before breaking the blind. Treatment assignment should remain blinded unless that knowledge is necessary to determine subject emergency medical care. The rationale for unblinding must be clearly explained in source documentation and on the electronic case report form (eCRF), along with the date on which the treatment assignment was obtained. The investigator is requested to contact the Gilead Medical Monitor promptly in case of any treatment unblinding.

Blinding of study treatment is critical to the integrity of this clinical study and therefore, if a subject's treatment assignment is disclosed to the investigator, the subject will have study treatment discontinued. All subjects will be followed until study completion unless consent to do so is specifically withdrawn by the subject.

Gilead Drug Safety and Public Health (DSPH) may independently unblind cases for expedited reporting of suspected unexpected serious adverse reactions (SUSARs).

## 5.2. Description and Handling of GS-9674 and PTM GS-9674

#### 5.2.1. Formulation

GS-9674 is supplied as 30 mg and 100 mg strength (as free form equivalent) tablets. The tablets contain GS-9674-02 PPD

GS-9674 30 mg tablets are round, plain-faced, film-coated orange tablets and GS-9674 100 mg tablets are capsule-shaped, plain-faced, film-coated orange tablets.

Placebo-to-match (PTM) GS-9674 tablets are identical in size, shape, color, and appearance to their corresponding strengths of active GS-9674 tablets. PTM GS-9674 tablets

# 5.2.2. Packaging and Labeling

GS-9674 tablets and PTM GS-9674 tablets are packaged in white, high-density polyethylene (HDPE) bottles. Each bottle contains 30 tablets, a silica gel desiccant, and polyester packing material. Each bottle is enclosed with a white, continuous thread, child-resistant, polypropylene screw cap with an induction-sealed, aluminum-faced liner.

Study drug to be distributed to centers in the US and other participating countries shall be labeled to meet applicable requirements of the United States Food and Drug Administration (FDA), EU Guideline to Good Manufacturing Practice - Annex 13 (Investigational Medicinal Products), and/or other local regulations.

## 5.2.3. Storage and Handling

GS-9674 tablets and PTM GS-9674 tablets should be stored at controlled room temperature until required for administration. Controlled room temperature is defined as 25°C (77°F); temperature excursions are permitted between 15°C and 30°C (59°F and 86°F). Storage conditions are specified on the label.

Until study drug tablets are dispensed to the subjects, all bottles of study drugs should be stored in a securely locked area, accessible only to authorized site personnel. To ensure the stability and proper identification, the drug products should not be stored in a container other than the container in which they were supplied. Consideration should be given to handling, preparation, and disposal through measures that minimize drug contact with the body. Appropriate precautions should be followed to avoid direct eye contact or exposure when handling GS-9674 tablets and PTM GS-9674 tablets.
# 5.3. Dosage and Administration of GS-9674/ PTM GS-9674

GS-9674 and GS-9674 PTM tablets will be provided by Gilead Sciences, Inc. In order to maintain the blind, each subject will be supplied with 2 bottles of tablets. One bottle will contain GS-9674 30 mg or PTM GS-9674 30 mg, the second bottle will contain GS-9674 100 mg or PTM GS-9674 100 mg. Dosing for each treatment group will be as follows:

- **Treatment Group A:** GS-9674 30 mg (1 x 30 mg tablet) + PTM GS-9674 100 mg (1 x PTM 100 mg tablet) administered orally once daily with food
- **Treatment Group B:** GS-9674 100 mg (1 x 100 mg tablet) + PTM GS-9674 30 mg (1 x PTM 30 mg tablet) administered orally once daily with food
- Treatment Group C: PTM GS-9674 30 mg (1 x PTM 30 mg tablet) + PTM GS-9674 100 mg (1 x PTM 100 mg tablet) administered orally once daily with food

The study drug dose should be taken at approximately the same time each day with food.

A dose will be considered missed if the subject cannot take the dose within 12 hours of their regular dosing time. If a subject misses a dose, the subject should take their next dose at the regular dosing time.

#### 5.4. Prior and Concomitant Medications

Concomitant use of certain medications or herbal/natural supplements with study drug may result in PK and/or PD interactions resulting in increases or decreases in exposure of study drug or these medications.

Concomitant medications taken within 30 days of screening through the follow-up visit need to be recorded in the source documents and electronic Case Report Forms (eCRFs).

Subjects with co-morbid diseases requiring medication(s) must be taking the medication(s) without a change in dose within 28 days of Baseline/Day 1.

GS-9674 increased atorvastatin exposure (39%) which does not necessitate a priori dose modification based on the LIPITOR $^{\otimes}$  USPI. Subjects taking atorvastatin with GS-9674 should be monitored as per label recommendations.

#### 5.5. Prohibited Medications

The following medications are prohibited from 28 days prior to Baseline/Day 1 up to and including the day of the last dose of study drug:

- Vitamin E
- Hematologic stimulating agents (eg, erythropoiesis-stimulating agents (ESAs); granulocyte colony stimulating factor (GCSF); thrombopoietin (TPO) mimetics)

- Chronic systemic immunosuppressants including, but not limited to, corticosteroids (prednisone equivalent of > 10 mg/day for > 2 weeks), azathioprine, or monoclonal antibodies (eg, infliximab). Use for <2 weeks total is allowed.
- Investigational agents or devices for any indication
- Concomitant use of certain medications or herbal/natural supplements (potent inhibitors of OATP or potent or moderate inducers of OATP, CYP2C8, P-gp, or CYP3A) with study drug(s) may result in PK interactions resulting in increases or decreases in exposure of study drug(s) or concomitant medications. Examples of representative medications which are prohibited from 28 days prior to Baseline/Day 1 up to and including the day of the last dose of study drug, are listed below in Table 5-1:

Table 5-1. List of Medications Prohibited and to be used with Caution

| Drug Class | Agents Disallowed | Use with Caution |
|---|---|---|
| Antibiotics | | Clarithromycin, Erythromycin |
| Acid Reducing Agents | H2-Receptor Antagonists <sup>a</sup> | Antacids <sup>b</sup> |
| Anticonvulsants <sup>c</sup> | Carbamazepine, Oxcarbazepine, Phenobarbital, Phenytoin | |
| Antimycobacterials <sup>c</sup> | Rifabutin, Rifapentine, Rifampin | |
| Endothelin Receptor<br>Antagonists | Bosentan | |
| Herbal/Natural<br>Supplements <sup>c</sup> | St. John's Wort, Echinaccea. Milk thistle (ie, silymarin), Chinese herb sho-saiko-to (or Xiao-Shai-Hu-Tang) | |
| Other <sup>c</sup> | Modafinil | |

a H2-Receptor Antagonists can be taken up to 3 days prior to study drug dosing.

Medications for disease conditions **excluded** from the protocol (eg, HIV-1, HBV, or HCV infection, active cancer, transplantation) are not listed under this prohibited medications section and are disallowed in the study.

## 5.6. Accountability for GS-9674/ PTM GS-9674

The investigator or designee (eg, pharmacist) is responsible for ensuring adequate accountability of all used and unused study drug bottles. This includes acknowledgement of receipt of each shipment of study drug (quantity and condition), subject dispensing records, and returned or destroyed study product. All used and unused study drug bottles dispensed to subjects must be returned to the site.

b Antacids that directly neutralize stomach pH (ie, Tums, Maalox) are permitted but may not be taken within 4 hours (before or after) study drug administration.

c May result in a decrease in the concentrations of study drug.

Study drug accountability records will be provided to each study site to:

- Record the date received and quantity of study drug bottles
- Record the date, subject number, subject initials, and the study drug bottle number dispensed
- Record the date, quantity of used and unused study drug returned, along with the initials of the person recording the information.

# 5.6.1. Investigational Medicinal Product Return or Disposal

Refer to Section 9.1.7 for instructions regarding study drug return or disposal.

## 6. STUDY PROCEDURES

The study procedures to be conducted for each subject enrolled in the study are presented in tabular form in Appendix 2 and described in the text that follows. Additional information is provided in the Study Reference Binder.

The investigator must document any deviation from protocol procedures and notify the sponsor or contract research organization (CRO).

# 6.1. Subject Enrollment and Treatment Assignment

It is the responsibility of the investigator to ensure that subjects are eligible to participate in the study prior to enrollment and throughout the study.

Documentation of the personally signed and dated informed consent of each subject, using the study-specific informed consent form (ICF), is required before initiating the screening process.

After written informed consent has been obtained and eligibility to participate established, investigative site personnel will obtain the subject's identification number and study drug assignment from the interactive web response system (IWRS).

# 6.2. Pretreatment Assessments – Screening Visit

Subjects will be screened within 4 weeks prior to randomization to determine eligibility for participation in the study. The screening period may be extended under special circumstances with the explicit approval of the Medical Monitor.

Screening labs may be repeated once within the screening period, prior to administration of study drug to rule out laboratory error, if any. This will be done at the discretion of the investigator and with prior approval of the Medical Monitor.

Subjects who fail to meet eligibility criteria may be rescreened once if there is a reasonable expectation that the subject will meet eligibility criteria after repeat screening.

Subjects should be <u>instructed to fast</u> (no food or drink, except water), starting from midnight (00:00) or earlier, as appropriate, on the evening prior to the Screening visit to ensure an approximate 8-hour fast prior to the fasted blood sample collection the next morning.

The following will be performed and documented at Screening:

- Obtain written informed consent before initiation of any screening procedures
- Review and record whether the subject meets inclusion and exclusion criteria
- Obtain screening number from IWRS

- Obtain medical history
- Complete physical examination
- Record vital signs, body weight, and height
- Obtain blood samples for:
  - Chemistry
  - Hematology
  - Coagulation Panel
  - Hemoglobin A1c
  - Biomarkers
  - HIV-1, HBV, and HCV Serology
  - Serum pregnancy test (only for female subjects of child bearing potential)
  - Serum FSH (only for some female subjects see Appendix 4)
- Conduct standard 12-Lead ECG
- Perform Ultrasound (if necessary) for confirmation of NAFLD
- Perform MRE and MRI-PDFF
- Urine drug screen for amphetamines, cocaine and opiates (ie, heroin, morphine)
- Record all concomitant medications that the subject has taken within 30 days prior to screening
- Record any serious adverse events and all adverse events related to protocol mandated procedures occurring after signing of the consent form.

Subjects meeting all of the inclusion criteria and none of the exclusion criteria will return to the clinic within 4 weeks of the start of screening for randomization into the study.

From the time of obtaining informed consent through the first administration of the study drug, record all serious adverse events (SAEs), as well as any adverse events related to protocol-mandated procedures on the adverse events electronic case report form (eCRF). All other untoward medical occurrences observed during the screening period, including exacerbation or changes in medical history are to be captured on the medical history eCRF. See Section 7 Adverse Events and Toxicity Management for additional details.

# 6.3. Baseline/Day 1 Randomization and Assessments

Subjects returning to the clinic for randomization at Baseline/Day 1 should be <u>instructed to fast</u> (no food or drink, except water), starting from midnight (00:00) or earlier, as appropriate, on the evening prior to the visit to ensure an approximate 8-hour fast prior to the blood sample collection under fasting condition the next morning.

After review of inclusion and exclusion criteria to confirm continued eligibility, subjects will be randomized to study drug assignment and receive their Subject Identification Number via the IWRS prior to their first dose of study drug.

The following will be performed and documented at the Baseline/Day 1 visit prior to dosing:

- QoL: general assessments (CLDQ, SF-36, and WPAI)
- QoL: pruritus assessments (VAS-itch and 5D-itch)

Note: It is recommended that QoL assessments be completed prior to any study procedures being performed and prior to the subject seeing a health care provider. Refer to the Study Reference Binder for guidance on QoL assessment administration.

- Symptom driven physical examination
- Record vital signs, waist circumference, and body weight

| | ~ | The second second | 1 | 1 1 | | 4 | 0 |
|---|----|-------------------|---|------|------|------|------|
| • | () | btain | h | lood | sami | nles | tor. |

| <u>2 5</u> | Chemistry |
|-------------|-------------------|
| <del></del> | Hematology |
| <u></u> 9 | Coagulation Panel |
| 1 | Lipid Profile |

- Hemoglobin A1c
- Biomarkers
- Single PD Sampling

\_\_ PPD

- Conduct standard 12-Lead ECG
- Perform FibroScan® (if available)

- Collect urine samples for:
  - Urine pregnancy test for females of child bearing potential only
  - Biomarker testing
- Collect stool sample for biomarker testing
- Dispense study drug and provide subject with instruction on appropriate dosing and administration;
- Record all concomitant medications that the subject has taken since the previous visit
- Record any serious adverse events and all adverse events occurring since the screening visit

Once all visit procedures have been completed, subjects will take their Baseline/Day 1 dose of study drug with food while at the investigative site.

Subjects will return to the investigative site at Week 1 (±3 days) for a mandatory safety visit. Then, starting at the Week 4 visit, subjects will have visits every 4 weeks up to the Week 24 visit.

#### **6.4.** Treatment Assessments

#### 6.4.1. Week 1

Subjects should be <u>instructed to fast</u> (no food or drink, except water), starting from midnight (00:00) or earlier, as appropriate, on the evening prior to the Week 1 visit to ensure an approximate 8-hour fast prior to the fasted blood sample collection the next morning.

Subjects should also be <u>instructed to HOLD their dose of study drug</u> on the day of their Week 1 visit until all visit procedures have been completed. The study drug dose should be taken with food after the visit.

During the Week 1 safety visit the following will be performed and documented (±3 days):

- QoL: pruritus assessments (VAS-itch and 5D-itch)
- Symptom driven physical examination
- Record vital signs and body weight
- Obtain blood samples for:
  - Chemistry
  - Hematology

- Coagulation Panel
- Lipid Profile
- Biomarkers
- Single PK and PD sampling
- Collect urine sample for biomarker testing
- Record all concomitant medications that the subject has taken since the previous visit
- Record any serious adverse events and all adverse events occurring since the previous visit

#### **6.4.2.** Week 4 Visit

Subjects should be <u>instructed to fast</u> (no food or drink, except water), starting from midnight (00:00) or earlier, as appropriate, on the evening prior to the Week 4 visit to ensure an approximate 8-hour fast prior to the fasted blood sample collection the next morning.

Subjects should also be <u>instructed to HOLD their dose of study drug</u> on the day of their Week 4 visit until all visit procedures have been completed. The study drug dose should be taken with food after the visit.

The following will be performed and documented at this visit ( $\pm 3$  days):

- QoL: pruritus assessments (VAS-itch and 5D-itch)
- Symptom driven physical examination
- Record vital signs and body weight
- Obtain blood samples for:
  - Chemistry
  - Hematology
  - Coagulation Panel
  - Lipid Profile
  - Biomarkers
  - Single PK and PD sampling

- Collect urine samples for:
  - Urine pregnancy test for females of child bearing potential only
  - Biomarker testing
- Dispense study drug
- Record all concomitant medications that the subject has taken since the previous visit
- Record any serious adverse events and all adverse events occurring since the previous visit

## 6.4.3. Week 8, 16, and 20 Visits

Subjects should be <u>instructed to fast</u> (no food or drink, except water), starting from midnight (00:00) or earlier, as appropriate, on the evening prior to the Weeks 8, 16, and 20 visits to ensure an approximate 8-hour fast prior to the fasted blood sample collection the next morning.

Subjects should also be <u>instructed to HOLD their dose of study drug</u> on the day of their Weeks 8, 16, and 20 visits until all visit procedures have been completed. The study drug dose should be taken with food after the visit.

The following will be performed and documented at these visits ( $\pm 3$  days):

- QoL: pruritus assessments (VAS-itch and 5D-itch)
- Symptom driven physical examination
- Record vital signs and body weight
- Obtain blood samples for:
  - Chemistry
  - Hematology
  - Coagulation Panel
  - Lipid Profile
  - Single PK and PD sampling
- Urine pregnancy test for females of child bearing potential only
- Dispense study drug
- Record all concomitant medications that the subject has taken since the previous visit
- Record any serious adverse events and all adverse events occurring since the previous visit

## 6.4.4. Week 12 Visit

Subjects should be <u>instructed to fast</u> (no food or drink, except water), starting from midnight (00:00) or earlier, as appropriate, on the evening prior to the Week 12 visit to ensure an approximate 8-hour fast prior to the fasted blood sample collection the next morning.

Subjects should also be <u>instructed to HOLD their dose of study drug</u> on the day of their Week 12 visit until all visit procedures have been completed. The study drug dose should be taken with food after the visit

The following will be performed and documented at this visit ( $\pm 7$  days):

- QoL: general assessments (CLDQ, SF-36, and WPAI)
- QoL: pruritus assessments (VAS-itch and 5D-itch)
- Symptom driven physical examination
- Record vital signs and body weight
- Obtain blood samples for:
  - Chemistry
  - Hematology
  - Coagulation Panel
  - Lipid Profile
  - Hemoglobin A1c
  - Biomarkers
  - Single PK and PD sampling
- Collect urine samples for:
  - Urine pregnancy test for females of child bearing potential only
  - Biomarker testing
- Conduct standard 12-Lead ECG
- Perform FibroScan® (if available)
- Perform MRE and MRI-PDFF

- Dispense study drug
- Record all concomitant medications that the subject has taken since the previous visit
- Record any serious adverse events and all adverse events occurring since the previous visit

# 6.4.5. Week 24 Visit

Subjects should be <u>instructed to fast</u> (no food or drink, except water), starting from midnight (00:00) or earlier, as appropriate, on the evening prior to the Week 24 visit to ensure an approximate 8-hour fast prior to the fasted blood sample collection the next morning.

Subjects should also be <u>instructed to HOLD their dose of study drug</u> on the day of their Week 24 visit until all visit procedures have been completed.

The following will be performed and documented at this visit ( $\pm 7$  days):

- QoL: general assessments (CLDQ, SF-36, and WPAI)
- QoL: pruritus assessments (VAS-itch and 5D-itch)
- Symptom driven physical examination
- Record vital signs, waist circumference, and body weight
- Obtain blood samples for:
  - Chemistry
  - Hematology
  - Coagulation Panel
  - Lipid Profile
  - Hemoglobin A1c
  - Biomarkers
  - Single PK and PD sampling
- Collect urine samples for:
  - Urine pregnancy test for females of child bearing potential only
  - Biomarker testing
- Conduct standard 12-Lead ECG
- Perform FibroScan® (if available)

- Perform MRE and MRI-PDFF
- Collect stool sample for biomarkers
- Record all concomitant medications that the subject has taken since the previous visit
- Record any serious adverse events and all adverse events occurring since the previous visit

Once all visit procedures have been completed, subjects will take their final dose of study drug while at the investigative site.

PPD

#### 6.4.6. Unscheduled Visits

Additional unscheduled assessments may be performed at the discretion of the investigator.

Subjects returning to the clinic for an unscheduled visit should be <u>instructed to fast</u> (no food or drink, except water), starting from midnight (00:00) or earlier, as appropriate, on the evening prior to the visit to ensure an approximate 8-hour fast prior to the blood sample collection under fasting condition the next morning.

Subjects should also be <u>instructed to HOLD their dose of study drug</u> on the day of an unscheduled visit until all visit procedures have been completed. The study drug dose should be taken with food after the visit.

At a minimum, the following will be performed and documented.

- Symptom driven physical examination
- Record body weight
- Obtain blood samples for:
  - Chemistry
  - Hematology
- Record all concomitant mediations that the subject has taken since the previous visit
- Record any serious adverse events and all adverse events occurring since the previous visit

If the Unscheduled visit is performed for the sole purpose of distribution of study drug, the assessments noted above do not need to be performed.

# 6.5. Follow-Up Visit

Subjects will return for a Follow-Up Visit four weeks after their last dose of study drug.

Subjects should be <u>instructed to fast</u> (no food or drink, except water), starting from midnight (00:00) or earlier, as appropriate, on the evening prior to the Follow-Up visit to ensure an approximate 8-hour fast prior to the blood sample collection under fasting condition the next morning.

The following will be performed and documented at this visit ( $\pm 5$  days):

- Symptom driven physical examination
- Record vital signs and body weight
- Obtain blood samples for:
  - Chemistry
  - Hematology
  - Coagulation Panel
- Urine pregnancy test for female subjects of child bearing potential only
- Record all concomitant medications that the subject has taken since the previous visit
- Record any serious adverse events and all adverse occurring since the previous visit

## 6.6. Assessments for Premature Discontinuation from Study

Subjects prematurely discontinuing from the study (for example, as a result of an AE), should have an Early Termination (ET) visit, if possible, and a Follow-Up visit 4 weeks after their last dose of study drug. The study assessments to be performed at the ET visit are the same as those performed at the Week 24 visit (refer to Section 6.4.5). The study assessments to be performed at the Follow-Up visit are listed in Section 6.5. The subject will then be withdrawn from the study.

If these visits are not possible or acceptable to the subject or investigator, the subject may be withdrawn from the study.

# 6.7. Criteria for Discontinuation of Study Treatment

Study medication may be discontinued in the following instances:

- Intercurrent illness that would, in the judgment of the investigator, affect assessments of
  clinical status to a significant degree. Following resolution of intercurrent illness, the subject
  may resume study dosing at the discretion of the investigator.
- Unacceptable toxicity, or toxicity that, in the judgment of the investigator, compromises the
  ability to continue study-specific procedures or is considered to not be in the subject's best
  interest
- Subject request to discontinue for any reason
- Subject noncompliance
- Pregnancy during the study (refer to Appendix 4)
- Sponsor discretion
- Discontinuation of the study at the request of Gilead, a regulatory agency or an institutional review board, independent ethics committee, or ethics committee (IRB/IEC/EC)

# 6.8. PK and PD Substudy Visits



# 6.9. Description of Assessments

## 6.9.1. Clinical Laboratory Analytes

#### Chemistry:

alanine aminotransferase (ALT), aspartate aminotransferase (AST), albumin, alkaline phosphatase (ALP), bicarbonate, blood urea nitrogen (BUN), calcium, chloride, creatinine, glucose, lactate dehydrogenase (LDH), magnesium, phosphorus, potassium, sodium, total and direct bilirubin, total protein, uric acid, gamma-glutamyl transferase (GGT). Also includes C-Peptide and Insulin for the Baseline/Day1, Weeks 4, 12, and 24 visits.

Creatinine clearance is calculated by the Cockcroft-Gault equation {Cockcroft et al 1976} using actual body weight (BW). The calculation will be performed by the central laboratory.

# Hematology:

Hematocrit (Hct), Hemoglobin (Hb), Platelet count, Red blood cell count (RBC), White blood cell count (WBC) with differential (absolute and percentage) including Lymphocytes, Monocytes, Neutrophils, Eosinophils, and Basophils and, Reticulocyte count and mean corpuscular volume (MCV).

### Coagulation Panel:

Prothrombin time (PT), partial thromboplastin time (PTT), and international normalized ratio (INR)

## Pregnancy Tests:

Serum  $\beta$ -hCG or urine  $\beta$ -hCG (if positive, requires immediate confirmation with Serum  $\beta$ -hCG)

## Additional Tests:

Lipid Profile, Hemoglobin A1c, HIV-1, HBV & HCV Serology, urine drug screen (for amphetamines, cocaine, opiates), creatine phosphokinase, and genomic sample collection.

#### Biomarker Tests:

CK18 (M30 and M65), FGF-19, C4, Apolipoprotein B (Apo B), metabolite profile, bile acids, stool microbiome, blood miRNA, NMR lipoprofile, free fatty acids, ELF™ Test, and FibroSURE/FibroTest®.

PPD

# Pharmacokinetic (PK) and Pharmacodynamic (PD) Assessments

Single PK and PD Sampling

Single PK and PD plasma samples will be collected and archived for 1) PK analysis of GS-9674, GS-716070 (metabolite of GS-9674), and other metabolites as applicable, 2) to measure the concentration of the PD biomarkers FGF19 and C4.

PK and PD Substudy

PPD

# 6.9.2. Medical History

Medical history, including details of illnesses and allergies, date(s) of onset, whether condition(s) is currently ongoing, and medication history, including nicotine and alcohol use, will be collected for all subjects during screening.

### 6.9.3. Physical Examination

A complete physical examination should include source documentation of general appearance, and the following body systems: head, neck, and thyroid; eyes, ears, nose, throat, mouth, and tongue; chest (excluding breasts); respiratory; cardiovascular; lymph nodes; abdomen; skin, hair, nails; musculoskeletal; neurological.

The focus of a symptom driven physical examination will be determined by the investigator based on subject complaint. For eg, if a subject complains of a cough, a lung exam should be performed. If consistent with pneumonia (rales/crackles on exam) then an AE would be documented.

Height, body weight, and hip circumference will be collected at specified time points.

## 6.9.4. Quality of Life (QoL) Assessments

It is recommended that these questionnaires be completed prior to the clinical and laboratory assessments. The subject should read the questionnaires by himself/herself and record the answers by himself/herself.

## 6.9.4.1. Chronic Liver Disease Questionnaire (CLDQ)

The CLDQ asks 29 questions related to liver disease to measure health related quality of life in subjects with chronic liver disease.

# 6.9.4.2. SF-36 Health Survey

The SF-36 Health Survey asks 36 questions to measure functional health and well-being from the subject's point of view and consists of eight health domains (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health). These health domain scales contribute to the physical health and mental health summary measures.

## 6.9.4.3. Work Productivity and Activity Impairment (WPAI)

The Work Productivity and Activity Impairment (WPAI) questionnaire asks 6 questions regarding the effect of NASH on a person's ability to work and perform regular activities.

#### 6.9.4.4. VAS-itch

The visual analogue scale (VAS)-itch is a tool for measuring the intensity of pruritus.

#### 6.9.4.5. 5-D itch

The 5-D itch is multidimensional measure of itching that allows changes in chronic pruritus to be detected over time. The questionnaire measures the degree, duration, direction, disability, and distribution of pruritus.

# 6.9.5. Electrocardiogram

Standard 12-lead electrocardiogram (ECG) assessments will be performed. The investigator will review the ECGs for any clinically significant abnormalities to ensure subject safety. Abnormal ECG findings that are considered clinically significant by the investigator and meet the definition of an AE should be reported and recorded in the AE eCRF page.

## 6.9.6. FibroScan®

Liver stiffness will be assessed by FibroScan<sup>®</sup>. It is required that each subject's FibroScan<sup>®</sup> assessments be done with the same type of probe at each study visit. If FibroScan<sup>®</sup> is not available at a site the test may be omitted.

Please refer to the Study Reference Binder for instructions on FibroScan® measurements.

## 6.9.7. MRE and MRI-PDFF

Liver stiffness will be assessed by MRE and the degree of steatosis will be measured by Magnetic Resonance Imaging-Proton Density Fat Fraction (MRI-PDFF). These assessments can occur sequentially.

The MRE and MRI-PDFF images will be analyzed by a central reader.

Please refer to the Study Reference Binder for MRE and MRI-PDFF imaging guidelines.

# 6.10. End of Study Definition

End of study is defined as when the last patient last visit (LPLV) for the Follow-Up visit (four weeks after their last dose of study drug) occurs, or the ET visit, whichever occurs later.

# 6.11. Post Study Care

No post study ongoing care will be provided.

## 7. ADVERSE EVENTS AND TOXICITY MANAGEMENT

# 7.1. Definitions of Adverse Events, Adverse Reactions, and Serious Adverse Events

#### 7.1.1. Adverse Events

An adverse event (AE) is any untoward medical occurrence in a clinical study subject administered a medicinal product, which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs may also include pre- or post-treatment complications that occur as a result of protocol specified procedures, overdose, drug abuse/misuse reports, or occupational exposure. Preexisting events that increase in severity or change in nature during or as a consequence of participation in the clinical study will also be considered AEs.

An AE does not include the following:

- Medical or surgical procedures such as surgery, endoscopy, tooth extraction, and transfusion. The condition that led to the procedure may be an adverse event and must be reported.
- Pre-existing diseases, conditions, or laboratory abnormalities present or detected before the Screening visit that do not worsen.
- Situations where an untoward medical occurrence has not occurred (eg, hospitalization for elective surgery, social and/or convenience admissions).
- Overdose without clinical sequelae (see Section 7.6.1).
- Any medical condition or clinically significant laboratory abnormality with an onset date before the consent form is signed and not related to a protocol-associated procedure is not an AE. It is considered to be pre-existing and should be documented on the medical history eCRF.

#### 7.1.2. Serious Adverse Events

A **serious adverse event** (SAE) is defined as an event that, at any dose, results in the following:

- Death
- Life-threatening (Note: The term "life-threatening" in the definition of "serious" refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if it were more severe.)
- In-patient hospitalization or prolongation of existing hospitalization

- Persistent or significant disability/incapacity
- A congenital anomaly/birth defect
- A medically important event or reaction: such events may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes constituting SAEs. Medical and scientific judgment must be exercised to determine whether such an event is a reportable under expedited reporting rules. Examples of medically important events include intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization; and development of drug dependency or drug abuse. For the avoidance of doubt, infections resulting from contaminated medicinal product will be considered a medically important event and subject to expedited reporting requirements.

# 7.1.3. Clinical Laboratory Abnormalities and Other Abnormal Assessments as Adverse Events or Serious Adverse Events

Laboratory abnormalities without clinical significance are not recorded as AEs or SAEs. However, laboratory abnormalities (eg, clinical chemistry, hematology, and urinalysis) that require medical or surgical intervention or lead to study drug interruption, modification, or discontinuation must be recorded as an AE, as well as an SAE, if applicable. In addition, laboratory or other abnormal assessments (eg, electrocardiogram, x-rays, vital signs) that are associated with signs and/or symptoms must be recorded as an AE or SAE if they meet the definition of an AE or SAE as described in Sections 7.1.1 and 7.1.2. If the laboratory abnormality is part of a syndrome, record the syndrome or diagnosis (eg, anemia), not the laboratory result (ie, decreased hemoglobin).

#### 7.2. Assessment of Adverse Events and Serious Adverse Events

The investigator or qualified subinvestigator is responsible for assessing AEs and SAEs for causality and severity, and for final review and confirmation of accuracy of event information and assessments.

# 7.2.1. Assessment of Causality for Study Drugs and Procedures

The investigator or qualified subinvestigator is responsible for assessing the relationship to GS-9674 therapy using clinical judgment and the following considerations:

- No: Evidence exists that the adverse event has an etiology other than the GS-9674. For SAEs, an alternative causality must be provided (eg, pre-existing condition, underlying disease, intercurrent illness, or concomitant medication).
- Yes: There is reasonable possibility that the event may have been caused by the study drug.

It should be emphasized that ineffective treatment should not be considered as causally related in the context of adverse event reporting.

The relationship to study procedures (eg, invasive procedures such as venipuncture or biopsy) should be assessed using the following considerations:

- No: Evidence exists that the adverse event has an etiology other than the study procedure.
- Yes: The adverse event occurred as a result of protocol procedures (eg, venipuncture)

# 7.2.2. Assessment of Severity

The severity grading of AEs will be assessed as Grade 1, 2, 3, 4, or 5 according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, which can be found at http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE\_4.03\_2010-06-14\_QuickReference\_8.5x11.pdf (Appendix 3).

For AEs associated with laboratory abnormalities, the event should be graded on the basis of the clinical severity in the context of the underlying conditions; this may or may not be in agreement with the grading of the laboratory abnormality.

The distinction between the seriousness and the severity of an adverse event should be noted. Severe is a measure of intensity; thus, a severe reaction is not necessarily a serious reaction. For example, a headache may be severe in intensity, but would not be classified as serious unless it met one of the criteria for serious events listed above.

# 7.3. Investigator Requirements and Instructions for Reporting Adverse Events and Serious Adverse Events to Gilead

Requirements for collection prior to study drug initiation:

After informed consent, but prior to initiation of study medication, the following types of events should be reported on the electronic case report form (eCRF): all SAEs and adverse events related to protocol-mandated procedures.

#### **Adverse Events**

Following initiation of study medication, collect all AEs, regardless of cause or relationship, until 30 days after last administration of GS-9674; AEs must be reported to the eCRF database as instructed.

All AEs should be followed up until resolution or until the adverse event is stable, if possible. Gilead Sciences may request that certain AEs be followed beyond the protocol defined follow up period.

#### **Serious Adverse Events**

All SAEs, regardless of cause or relationship, that occur after the subject first consents to participate in the study (ie, signs the informed consent) and throughout the duration of the study, including the protocol-required post treatment follow-up period, must be reported to the eCRF database and Gilead Drug Safety and Public Health (DSPH) as instructed. This also includes any SAEs resulting from protocol-associated procedures performed after informed consent is signed.

Any SAEs and deaths that occur after the post treatment follow-up visit but within 30 days of the last dose of GS-9674, regardless of causality, should also be reported.

Investigators are not obligated to actively seek SAEs after the protocol defined follow up period; however, if the investigator learns of any SAEs that occur after study participation has concluded and the event is deemed relevant to the use of study drug, he/she should promptly document and report the event to Gilead DSPH.

• All AEs and SAEs will be recorded in the eCRF database within the timelines outlined in the eCRF completion guideline.

Electronic Serious Adverse Event (eSAE) Reporting Process

- Site personnel record all SAE data in the eCRF database and from there transmit the SAE information to Gilead DSPH within 24 hours of the investigator's knowledge of the event. Detailed instructions can be found in the eCRF completion guidelines.
- If for any reason it is not possible to record the SAE information electronically, ie, the eCRF database is not functioning, record the SAE on the paper serious adverse event reporting form (see Study Reference Binder) and submit within 24 hours to:

Gilead DSPH: Fax: +1 (650) 522-5477

Email: Safety FC@gilead.com

- As soon as it is possible to do so, any SAE reported via paper must be transcribed into the eCRF Database according to instructions in the eCRF completion guidelines.
- If an SAE has been reported via a paper form because the eCRF database has been locked, no further action is necessary.
- For fatal or life-threatening events, copies of hospital case reports, autopsy reports, and other documents are also to be submitted by e-mail or fax when requested and applicable.
   Transmission of such documents should occur without personal subject identification, maintaining the traceability of a document to the subject identifiers.
- Additional information may be requested to ensure the timely completion of accurate safety reports.
- Any medications necessary for treatment of the SAE must be recorded onto the concomitant medication section of the subject's eCRF and the event description section of the SAE form.

# 7.4. Gilead Reporting Requirements

Depending on relevant local legislation or regulations, including the applicable US FDA Code of Federal Regulations, the EU Clinical Trials Directive (2001/20/EC) and relevant updates, and other country-specific legislation or regulations, Gilead may be required to expedite to worldwide regulatory agencies reports of SAEs, serious adverse drug reactions (SADRs), or suspected unexpected serious adverse reactions (SUSARs). In accordance with the EU Clinical Trials Directive (2001/20/EC), Gilead or a specified designee will notify worldwide regulatory agencies and the relevant IEC in concerned Member States of applicable SUSARs as outlined in current regulations.

Assessment of expectedness for SAEs will be determined by Gilead using reference safety information specified in the investigator's brochure or relevant local label as applicable.

All investigators will receive a safety letter notifying them of relevant SUSAR reports associated with any study drug. The investigator should notify the IRB or IEC of SUSAR reports as soon as is practical, where this is required by local regulatory agencies, and in accordance with the local institutional policy.

To minimize the possibility of exposing study subjects to unusual risk, the safety information from this study will also be reviewed periodically by an independent Data Monitoring Committee (DMC). The DMC may have access to partially blinded or unblinded data and will make recommendations regarding the study according to the DMC charter. See Section 8.11 for additional details regarding the DMC.

## 7.5. Toxicity Management

Observation for Drug Induced Liver Injury (DILI):

Although subjects enrolled in this study will have baseline liver disease, their hepatic function should not be significantly impaired. However, at baseline, some may have liver biochemistry levels above the upper limit of normal (ULN). Baseline values for liver tests (ALT, AST, total bilirubin, and ALP) will be determined by averaging the values obtained at screening and baseline/Day1.

For subjects with ALT and AST below ULN at study start, close observation for DILI (as described below) will be performed in subjects with any of the following criteria (all labs confirmed by repeat testing):

- ALT or AST > 3 x ULN at any time
- Total bilirubin > 2 x ULN
- $ALP > 3 \times ULN$
- INR >1.5 (except for subjects on anticoagulant therapy)

• Clinical signs or symptoms that are, in the opinion of the investigator, consistent with hepatitis (such as right upper quadrant discomfort, fever, nausea, vomiting, jaundice, rash, or eosinophilia > 5%)

For subjects with ALT or AST between 1 and 5 x ULN at study start, close observation for DILI (as described below) will be performed in subjects with any of the following criteria (all labs confirmed by repeat testing):

- ALT or AST > 2 x baseline at any time
- Total bilirubin > 2 x ULN
- Alkaline phosphatase > 3 x ULN
- INR >1.5 (except for subjects on anticoagulant therapy)
- Clinical signs or symptoms that are, in the opinion of the investigator, consistent with hepatitis (such as right upper quadrant discomfort, fever, nausea, vomiting, jaundice, rash, or eosinophilia > 5%).

#### Close observation includes:

- Repeating liver biochemistries (ALT, AST, ALP, total bilirubin, INR) and obtaining creatine phosphokinase (CPK) levels within 48 hours
- Obtaining a more detailed history of symptoms and prior or concurrent disease
- Obtaining a history of concomitant drug use (including nonprescription medications and herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets
- Obtaining a history of exposure to environmental chemical agents
- Ruling out other causes of liver disease as needed (obtain viral hepatitis panel, imaging for evaluation of biliary tract disease, etc. if required in the opinion of the primary investigator)
- Continue to monitor liver biochemistries twice weekly. Frequency can decrease to once a
  week or less if abnormalities stabilize or study drug has been discontinued and subject is
  asymptomatic

During a period of close observation, study drug can be continued, if desired, at the discretion of the Gilead Medical Monitor and the principal investigator during the DILI evaluation.


However, for all subjects, study drug should be withheld if any of the following criteria are met:

- ALT or AST > 5 x baseline
- ALT or AST >10 x ULN
- ALT or AST >3 x baseline with 1 or more of the following:
  - Total bilirubin > 2 x ULN or 1.5 x baseline
  - INR >1.5 (except for subjects on anticoagulant therapy)
  - Appearance of clinical signs or symptoms that are, in the opinion of the investigator, consistent with drug-induced hepatotoxicity
- ALT or AST > baseline with any 2 or more of the following:
  - Total bilirubin > 2 x ULN or 1.5 x baseline
  - INR >1.5 (except for subjects on anticoagulant therapy)
  - Appearance of clinical signs or symptoms that are, in the opinion of the investigator, consistent with drug-induced hepatotoxicity

#### **AND**

- No other cause for the combination of laboratory abnormalities is immediately apparent (eg, prolonged INR with warfarin use) important potential causes or contributors to abnormal AST/ALT or total bilirubin values include, but are not limited to:
  - Obstructive gall bladder or bile duct disease
  - Viral or alcoholic hepatitis (eg, hepatitis A/B/C/D/E, Epstein-Barr virus, cytomegalovirus, herpes simplex virus, varicella)
  - Autoimmune hepatitis
  - Concomitant administration of other hepatotoxins, including excessive doses of acetaminophen, drugs that inhibit bilirubin glucuronidation (eg, indinavir, atazanavir, irinotecan), or herbal or dietary supplements
  - Hypoxic or ischemic hepatopathy or congestive hepatopathy in association with significant right-sided heart failure
  - Wilson disease
  - Progression of malignancy involving the liver (note that metastatic disease to the liver, by itself, should not be used as an explanation for significant AST/ALT elevations)


If study drugs are withheld, they may be reintroduced with approval from the Medical Monitor if another etiology for elevated liver tests is present. Study drug must be discontinued if close monitoring of a patient for DILI is not possible, or if total bilirubin, ALT or AST elevation recurs following re-challenge with study drug.

Treatment-emergent toxicities will be noted by the investigator and brought to the attention of the Medical Monitor. Whether or not considered treatment-related, all subjects experiencing AEs must be monitored periodically until symptoms subside, any abnormal laboratory values have resolved or returned to baseline levels or they are considered irreversible, or until there is a satisfactory explanation for the changes observed.

- Other than in the case of the liver enzymes noted above, Grade 3 or 4 clinically significant laboratory AEs should be confirmed by repeat testing as soon as practical to do so, and preferably within 3 calendar days of receipt of the original test results.
- For AEs associated with laboratory abnormalities, the event should be graded on the basis of the clinical severity in the context of the underlying conditions; this may or may not be in agreement with the grading of the laboratory abnormality.
- Any questions regarding toxicity management should be directed to the Medical Monitor.

## 7.6. Special Situations Reports

## 7.6.1. Definitions of Special Situations

Special situation reports include all reports of medication error, abuse, misuse, overdose, reports of AEs associated with product complaints, occupational exposure with an AE, pregnancy reports regardless of an associated AE, and AE in an infant following exposure from breastfeeding.

Medication error is any unintentional error in the prescribing, dispensing, or administration of a medicinal product while in the control of the health care provider, subject, or consumer.

Abuse is defined as persistent or sporadic intentional excessive use of a medicinal product by a subject.

Misuse is defined as any intentional and inappropriate use of a medicinal product that is not in accordance with the protocol instructions or the local prescribing information.

An overdose is defined as an accidental or intentional administration of a quantity of a medicinal product given per administration or cumulatively which is above the maximum recommended dose as per protocol or in the product labeling (as it applies to the daily dose of the subject in question). In cases of a discrepancy in drug accountability, overdose will be established only when it is clear that the subject has taken the excess dose(s). Overdose cannot be established when the subject cannot account for the discrepancy except in cases in which the investigator has reason to suspect that the subject has taken the additional dose(s).

Product complaint is defined as complaints arising from potential deviations in the manufacture, packaging, or distribution of the medicinal product.

Occupational exposure is defined as exposure to a medicinal product as a result of one's professional or non-professional occupation.

# 7.6.2. Instructions for Reporting Special Situations

## 7.6.2.1. Instructions for Reporting Pregnancies

The investigator should report pregnancies in female study subjects that are identified after initiation of study medication and throughout the study, including the post study drug follow-up period, to Gilead DSPH using the pregnancy report form within 24 hours of becoming aware of the pregnancy.

Refer to Section 7.3 and the eCRF completion guidelines for full instructions on the mechanism of pregnancy reporting.

The pregnancy itself is not considered an AE nor is an induced elective abortion to terminate a pregnancy without medical reasons.

Any premature termination of pregnancy (eg, a spontaneous abortion, an induced therapeutic abortion due to complications or other medical reasons) must be reported within 24 hours as an SAE. The underlying medical reason for this procedure should be recorded as the AE term.

A spontaneous abortion is always considered to be an SAE and will be reported as described in Sections 7.1.1 and 7.1.2. Furthermore, any SAE occurring as an adverse pregnancy outcome post study must be reported to Gilead DSPH.

The subject should receive appropriate monitoring and care until the conclusion of the pregnancy. The outcome should be reported to Gilead DSPH using the pregnancy outcome report form. If the end of the pregnancy occurs after the study has been completed, the outcome should be reported directly to Gilead DSPH. Gilead DSPH contact information is as follows: Email: Safety FC@gilead.com and Fax: +1 (650) 522-5477.

Pregnancies of female partners of male study subjects exposed to Gilead or other study drugs must also be reported and relevant information should be submitted to Gilead DSPH using the pregnancy and pregnancy outcome forms within 24 hours. Monitoring of the subject should continue until the conclusion of the pregnancy. If the end of the pregnancy occurs after the study has been completed, the outcome should be reported directly to Gilead DSPH, fax number +1 650 522-5477 or email Safety FC@gilead.com.

Refer to Appendix 4 for Pregnancy Precautions, Definition for Female of Childbearing Potential, and Contraceptive Requirements.

# 7.6.2.2. Reporting Other Special Situations

All other special situation reports must be reported on the special situations report form and forwarded to Gilead DSPH within 24 hours of the investigator becoming aware of the situation. These reports must consist of situations that involve study drug and/or Gilead concomitant medications, but do not apply to non-Gilead concomitant medications.

Special situations involving non-Gilead concomitant medications does not need to be reported on the special situations report form; however, for special situations that result in AEs due to a non-Gilead concomitant medication, the AE should be reported on the AE form.

Any inappropriate use of concomitant medications prohibited by this protocol should not be reported as "misuse," but may be more appropriately documented as a protocol deviation.

Refer to Section 7.3 and the eCRF completion guidelines for full instructions on the mechanism of special situations reporting.

All clinical sequelae in relation to these special situation reports will be reported as AEs or SAEs at the same time using the AE eCRF and/or the SAE report form. Details of the symptoms and signs, clinical management, and outcome will be reported, when available.

# 8. STATISTICAL CONSIDERATIONS

Details will be provided in the statistical analysis plan (SAP).

# 8.1. Analysis Objectives and Endpoints

# 8.1.1. Analysis Objectives

The **primary objective** of this study is as follows:

• To evaluate the safety and tolerability of GS-9674 in subjects with NASH.

The **exploratory objectives** of this study are as follows:



# 8.1.2. Primary Endpoint

The primary endpoint is the safety of GS-9674 in subjects with NASH. Safety endpoints include adverse events and laboratory evaluations.

# 8.1.3. Exploratory Efficacy Endpoints



## 8.2. Analysis Conventions

All individual subject data will be listed as measured. All statistical summaries and analyses will be performed using SAS® software (SAS Institute, Cary, North Carolina, USA).

# 8.2.1. Analysis Sets

# 8.2.1.1. Efficacy

The primary analysis set for efficacy analysis is defined as the Full Analysis Set (FAS), which includes all subjects who were randomized into the study and received at least 1 dose of study drug.

Subjects who receive study drug other than that to which they were assigned for the entire duration of treatment, will be analyzed according to the treatment group they were randomized to.

## 8.2.1.2. Safety

The primary analysis set for safety analyses is defined as all subjects who received at least one dose of study drug. Subjects who receive study drug other than that to which they were assigned for the entire duration of treatment, will be analyzed according to the study drug received.

All data collected during treatment plus 30 days after last dose of study drug will be included in the safety summaries.

#### 8.2.1.3. Pharmacokinetics

There are two pharmacokinetic analysis sets: 1) The PK Analysis Set which includes concentration data from the single samples drawn at each visit PPD

The PK Analysis Set will include all enrolled or randomized subjects who took at least one dose of study drug and for whom concentration data of analytes GS-9674 (and its metabolites as applicable) are available. The PK Analysis Set will be used for analyses of population PK.

PPD

#### 8.2.1.4. Pharmacodynamics

There are two pharmacodynamic analysis sets: 1) The PD Analysis Set which includes concentration data from the single samples drawn at each visit PPD

The PD Analysis Set will include all enrolled or randomized subjects who took at least one dose of study drug and for whom concentration data of FGF19, C4, and bile acids are available. The PD Analysis Set may be used for descriptive and/or population based PD analyses as applicable.

PPD

#### 8.2.1.5. Biomarkers

The Biomarker Analysis Set will include data from subjects in the Safety Analysis Set who have the necessary baseline and on-study measurements to provide interpretable results for the specific parameters of interest.

## 8.2.2. Interim Analysis

An administrative interim analysis will be performed after all subjects finish 12 weeks of treatment

## 8.3. Data Handling Conventions

Missing data can have an impact on the interpretation of the study data. In general, values for missing data will not be imputed.

Where appropriate, safety data for subjects that did not complete the study will be included in summary statistics. For example, if a subject received study medication, the subject will be included in a summary of adverse events according to the treatment received; otherwise, if the subject is not dosed then they will be excluded from the summary. If safety laboratory results for a subject are missing for any reason at a time point, the subject will be excluded from the calculation of summary statistics for that time point. If the subject is missing a pre-dose value, then the subject will be excluded from the calculation of summary statistics for the pre-dose value and the change from pre-dose values.

Values for missing safety laboratory data will not be imputed; however, a missing baseline result will be replaced with a screening result, if available. If no pre-treatment laboratory value is available, the baseline value will be assumed to be normal (ie, no grade [Grade 0]) for the summary of graded laboratory abnormalities.

Values for missing vital signs data will not be imputed; however, a missing baseline result will be replaced with a screening result, if available.

## 8.4. Demographic Data and Baseline Characteristics

Demographic and baseline measurements will be summarized using standard descriptive methods.

Demographic summaries will include sex, race/ethnicity, and age.

Baseline data will include a summary of body weight, height, body mass index, and randomization stratification group (presence or absence of diabetes) and other disease characteristic variables.

## 8.5. Efficacy Analysis

The biological activity of GS-9674 will be evaluated using radiologic endpoints and biomarker variables. PPD

# 8.6. Safety Analysis

All safety data collected on or after the date that GS-9674 was first dispensed up to the date of last dose of GS-9674 plus 30 days will be summarized by treatment group. Data for the pretreatment and follow-up periods will be included in data listings.

# 8.6.1. Extent of Exposure

Data for a subject's extent of exposure to GS-9674 will be generated from the study drug administration eCRF. Exposure data will be summarized by treatment group.

#### **8.6.2.** Adverse Events

Clinical and laboratory adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). System Organ Class (SOC), High-Level Group Term (HLGT), High-Level Term (HLT), Preferred Term (PT), and Lower-Level Term (LLT) will be attached to the clinical database. Adverse event severity will be graded using the CTCAE Version 4 03

Events will be summarized on the basis of the date of onset for the event. A treatment-emergent adverse event (TEAE) will be defined as 1 or both of the following:

- Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug.
- Any AEs leading to premature discontinuation of study drug.

Summaries (number and percentage of subjects) of TEAEs by SOC and PT will be provided. Treatment-emergent AEs will also be summarized by relationship to study drug and severity. In addition, TEAEs leading to premature discontinuation of study drug and study will be summarized and listed

All AEs collected during the course of the study will be presented in data listings with a field for treatment-emergent event (yes/no).

# 8.6.3. Laboratory Evaluations

Selected laboratory data will be summarized (n, mean, SD, Median, Q1, Q3, minimum, and maximum) by treatment group and study visit along with the corresponding change from baseline values.

Graded laboratory abnormalities will be defined using the grading scheme in the CTCAE Version 4.03 (Appendix 3). Grading of laboratory abnormalities for analysis purposes will be performed by the central laboratory.

Incidence of treatment-emergent laboratory abnormalities, defined as values that increase at least 1 toxicity grade from baseline at any time post baseline up to and including the date of last dose

of study drug plus 30 days will be summarized by treatment group. If baseline data are missing, then any graded abnormality (ie, at least a Grade 1) will be considered treatment emergent.

# 8.6.4. Other Safety Evaluations

Summary statistics for the 12-lead ECGs performed at Baseline/Day 1, Week 12, and Week 24, will be generated.

# 8.7. Pharmacokinetic Analysis

Plasma concentrations and PK parameters (eg, AUC<sub>tau</sub>, C<sub>max</sub> and C<sub>tau</sub>) will be listed and summarized as appropriate for GS-9674 (and its metabolites as applicable) using descriptive statistics.

Details of the analysis plan will be provided in the Pharmacokinetic Reporting and Analysis Plan.

# 8.8. Pharmacodynamic Analysis

Primary PD parameters (AUC<sub>partial</sub>, C<sub>max</sub>, C<sub>min</sub> as applicable) of FGF19 and C4 will be listed and summarized as appropriate for GS-9674 using descriptive statistics.

Details of the analysis plan will be provided in the Pharmacodynamics Reporting and Analysis Plan.

# 8.9. Biomarker Analysis

Descriptive statistics of biomarker expression and change from baseline will be provided at each sampling time by treatment. Point estimates and 95% confidence intervals may be calculated.



# 8.10. Sample Size

Due to the exploratory nature of this study, no formal power calculations were used to determine sample size. The number of subjects was chosen based on clinical experience with other similar proof of concept studies. However, assuming that 4% of subjects in the placebo arm (N=25) and 32% in the GS-9674 100 mg arm (N=50) have a  $\geq$  30% reduction in MRI-PDFF at Week 24, this sample size will provide 80% power to detect the difference based on a two-sided Fisher's exact test at a significance level of 0.05.

# 8.11. Data Monitoring Committee

An independent, external data monitoring committee (DMC) that consists of two hepatologists and a PhD statistician will review the progress of the study and perform reviews of safety data. The DMC will convene once 20 subjects have been enrolled and will meet every 3 to 4 months thereafter to monitor the study for safety events. The DMC will meet on an ad hoc basis if there are at least 3 Grade ≥ 3 serious, treatment-related Common Terminology Criteria for Adverse Events (CTCAE) observed in the study. In the event of two similar Grade 4-CTCAE treatment-related adverse events or one Grade 5-CTCAE treatment-related adverse event, the DMC will review the data and advise the sponsor regarding stopping or continuing the study. The DMC will provide recommendation to Gilead whether the nature, frequency, and severity of adverse effects associated with study treatment warrant the early termination of the study in the best interests of the participants, whether the study should continue as planned, or the study should continue with modifications. The DMC may also provide recommendations as needed regarding study design.

The DMC's specific activities will be defined by a mutually agreed charter, which will define the DMC's membership, conduct, and meeting schedule.

While the DMC will be asked to advise Gilead regarding future conduct of the study, including possible early study termination, Gilead retains final decision-making authority on all aspects of the study.

## 9. RESPONSIBILITIES

# 9.1. Investigator Responsibilities

## 9.1.1. Good Clinical Practice

The investigator will ensure that this study is conducted in accordance with the principles of the Declaration of Helsinki, International Conference on Harmonisation (ICH) guidelines, or with the laws and regulations of the country in which the research is conducted, whichever affords the greater protection to the study subject. These standards are consistent with the European Union Clinical Trials Directive 2001/20/EC and Good Clinical Practice Directive 2005/28/EC.

The investigator will ensure adherence to the basic principles of Good Clinical Practice, as outlined in 21 CFR 312, subpart D, "Responsibilities of Sponsors and Investigators," 21 CFR, part 50, 1998, and 21 CFR, part 56, 1998.

The investigator and all applicable subinvestigators will comply with 21 CFR, Part 54, 1998, providing documentation of their financial interest or arrangements with Gilead, or proprietary interests in the investigational drug under study. This documentation must be provided prior to the investigator's (and any subinvestigator's) participation in the study. The investigator and subinvestigator agree to notify Gilead of any change in reportable interests during the study and for 1 year following completion of the study. Study completion is defined as the date when the last subject completes the protocol-defined activities.

# 9.1.2. Institutional Review Board (IRB)/Independent Ethics Committee (IEC)/ Ethics Committee (EC) Review and Approval

The investigator (or sponsor as appropriate according to local regulations) will submit this protocol, informed consent form, and any accompanying material to be provided to the subject (such as advertisements, subject information sheets, or descriptions of the study used to obtain informed consent) to an IRB/IEC/EC. The investigator will not begin any study subject activities until approval from the IRB/IEC/EC has been documented and provided as a letter to the investigator.

Before implementation, the investigator will submit to and receive documented approval from the IRB/IEC/EC any modifications made to the protocol or any accompanying material to be provided to the subject after initial IRB/IEC/EC approval, with the exception of those necessary to reduce immediate risk to study subjects.

#### 9.1.3. Informed Consent

The investigator is responsible for obtaining written informed consent from each individual participating in this study after adequate explanation of the aims, methods, objectives, and potential hazards of the study and before undertaking any study-related procedures. The investigator must use the most current IRB/IEC/EC-approved consent form for documenting
written informed consent. Each informed consent (or assent as applicable) will be appropriately signed and dated by the subject or the subject's legally authorized representative and the person conducting the consent discussion, and also by an impartial witness if required by the IRB/IEC/EC or local requirements. The consent form will inform subjects about genomic testing and sample retention.

# 9.1.4. Confidentiality

The investigator must assure that subjects' anonymity will be strictly maintained and that their identities are protected from unauthorized parties. Only subject initials, date of birth, another unique identifier (as allowed by local law) and an identification code will be recorded on any form or biological sample submitted to the Sponsor, IRB/IEC/EC or laboratory. Laboratory specimens must be labeled in such a way as to protect subject identity while allowing the results to be recorded to the proper subject. Refer to the Central Laboratory Services Manual for specific laboratory instructions. NOTE: The investigator must keep a screening log showing codes, names, and addresses for all subjects screened and for all subjects enrolled in the study. Subject data will be processed in accordance with all applicable regulations.

The investigator agrees that all information received from Gilead, including but not limited to the investigator brochure, this protocol, eCRF, the study drug, and any other study information, remain the sole and exclusive property of Gilead during the conduct of the study and thereafter. This information is not to be disclosed to any third party (except employees or agents directly involved in the conduct of the study or as required by law) without prior written consent from Gilead. The investigator further agrees to take all reasonable precautions to prevent the disclosure by any employee or agent of the study site to any third party or otherwise into the public domain.

# 9.1.5. Study Files and Retention of Records

The investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented and the study data to be subsequently verified. These documents should be classified into at least the following two categories: (1) investigator's study file, and (2) subject clinical source documents.

The investigator's study file will contain the protocol/amendments, CRF and query forms, IRB/IEC/EC and governmental approval with correspondence, informed consent, drug records, staff curriculum vitae and authorization forms, and other appropriate documents and correspondence.

The required source data should include sequential notes containing at least the following information for each subject:

- Subject identification (name, date of birth, gender);
- Documentation that subject meets eligibility criteria, ie, history, physical examination, and confirmation of diagnosis (to support inclusion and exclusion criteria);

- Documentation of the reason(s) a consented subject is not enrolled;
- Participation in study (including study number);
- Study discussed and date of informed consent;
- Dates of all visits;
- Documentation that protocol specific procedures were performed;
- Results of efficacy parameters, as required by the protocol;
- Start and end date (including dose regimen) of GS-9674, including dates of dispensing and return;
- Record of all adverse events and other safety parameters (start and end date, and including causality and severity);
- Concomitant medication (including start and end date, dose if relevant; dose changes);
- Date of study completion and reason for early discontinuation, if it occurs.

All clinical study documents must be retained by the investigator until at least 2 years or according to local laws, whichever is longer, after the last approval of a marketing application in an ICH region (ie, United States, Europe, or Japan) and until there are no pending or planned marketing applications in an ICH region; or, if no application is filed or if the application is not approved for such indication, until 2 years after the investigation is discontinued and regulatory authorities have been notified. Investigators may be required to retain documents longer if specified by regulatory requirements, by local regulations, or by an agreement with Gilead. The investigator must notify Gilead before destroying any clinical study records.

Should the investigator wish to assign the study records to another party or move them to another location, Gilead must be notified in advance.

If the investigator cannot provide for this archiving requirement at the study site for any or all of the documents, special arrangements must be made between the investigator and Gilead to store these records securely away from the site so that they can be returned sealed to the investigator in case of an inspection. When source documents are required for the continued care of the subject, appropriate copies should be made for storage away from the site.

# 9.1.6. Case Report Forms

For each subject consented, an electronic case report form (eCRF) will be completed by an authorized study staff member whose training for this function is documented according to study procedures. eCRF should be completed on the day of the subject visit to enable the sponsor to perform central monitoring of safety data. The Eligibility Criteria eCRF should be completed

only after all data related to eligibility have been received. Subsequent to data entry, a study monitor will perform source data verification within the electronic data capture (EDC) system. Original entries as well as any changes to data fields will be stored in the audit trail of the system. Prior to database lock (or any interim time points as described in the clinical data management plan), the investigator will use his/her log in credentials to confirm that the forms have been reviewed, and that the entries accurately reflect the information in the source documents. The eCRF capture the data required per the protocol schedule of events and procedures. System-generated or manual queries will be issued to the investigative site staff as data discrepancies are identified by the monitor or internal Gilead staff, who routinely review the data for completeness, correctness, and consistency. The site coordinator is responsible for responding to the queries in a timely manner, within the system, either by confirming the data as correct or updating the original entry, and providing the reason for the update (eg, data entry error). At the conclusion of the study, Gilead will provide the site with a read-only archive copy of the data entered by that site. This archive must be stored in accordance with the records retention requirements outlined in Section 9.1.5.

# 9.1.7. Investigational Medicinal Product Accountability and Return

Where possible, study drug should be destroyed at the site. If the site does not have acceptable procedures in place for drug destruction, arrangements will be made between the site and Gilead Sciences (or Gilead Sciences' representative) for return of unused study drug supplies. The study monitor will provide instructions for return.

The study monitor will evaluate each study center's study drug disposal procedures and provide appropriate instruction for destruction of unused study drug supplies. If the site has an appropriate standard operating procedure (SOP) for drug destruction as determined by Gilead QA, the site may destroy used (empty or partially empty) and unused study drug supplies in accordance with that site's approved SOP. A copy of the site's approved SOP will be obtained for central files

If study drug is destroyed on site, the investigator must maintain accurate records for all study drug destroyed. Records must show the identification and quantity of each unit destroyed, the method of destruction, and the person who disposed of the study drug. Upon study completion, copies of the study drug accountability records must be filed at the site. Another copy will be returned to Gilead. Refer to the Pharmacy Binder for study drug disposal/return instructions.

The study monitor will review study drug supplies and associated records at periodic intervals.

# 9.1.8. Inspections

The investigator will make available all source documents and other records for this study to Gilead's appointed study monitors, the IRB/IEC/EC, or to regulatory authority or health authority inspectors.

# 9.1.9. Protocol Compliance

The investigator is responsible for ensuring the study is conducted in accordance with the procedures and evaluations described in this protocol.

# 9.2. Sponsor Responsibilities

#### 9.2.1. Protocol Modifications

Protocol modifications, except those intended to reduce immediate risk to study subjects, may be made only by Gilead. The investigator must submit all protocol modifications to the IRB/IEC/EC in accordance with local requirements and receive documented IRB/IEC/EC approval before modifications can be implemented.

# 9.2.2. Study Report and Publications

A clinical study report (CSR) will be prepared and provided to the regulatory agencies. Gilead will ensure that the report meets the standards set out in the ICH Guideline for Structure and Content of Clinical Study Reports (ICH E3). Note that an abbreviated report may be prepared in certain cases.

Investigators in this study may communicate, orally present, or publish in scientific journals or other scholarly media only after the following conditions have been met: the results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form or the study has been completed at all study sites for at least 2 years.

The investigator will submit to Gilead any proposed publication or presentation along with the respective scientific journal or presentation forum at least 30 days before submission of the publication or presentation.

No such communication, presentation, or publication will include Gilead's confidential information (see Section 9.1.4).

The investigator will comply with Gilead's request to delete references to its confidential information (other than the study results) in any paper or presentation and agrees to withhold publication or presentation for an additional 60 days in order to obtain patent protection if deemed necessary.

#### 9.3. Joint Investigator/Sponsor Responsibilities

# 9.3.1. Payment Reporting

Investigators and their study staff may be asked to provide services performed under this protocol, eg, attendance at Investigator's Meetings. If required under the applicable statutory and regulatory requirements, Gilead will capture and disclose to Federal and State agencies any

expenses paid or reimbursed for such services, including any clinical study payments, meal, travel expenses or reimbursements, consulting fees, and any other transfer of value.

# 9.3.2. Access to Information for Monitoring

In accordance with regulations and guidelines, the study monitor must have direct access to the investigator's source documentation in order to verify the accuracy of the data recorded in the eCRF.

The monitor is responsible for routine review of the eCRF at regular intervals throughout the study to verify adherence to the protocol and the completeness, consistency, and accuracy of the data being entered on them. The monitor should have access to any subject records needed to verify the entries on the eCRF. The investigator agrees to cooperate with the monitor to ensure that any problems detected through any type of monitoring (central, on site) are resolved.

# 9.3.3. Monitoring and Oversight of Biomarker Specimens

Biomarker research specimens will be tracked in a manner consistent with Good Clinical Practice by a quality-controlled, auditable, and appropriately validated laboratory information management system, to ensure compliance with data confidentiality as well as adherence to authorized use of specimens as specified in this protocol and in the Informed Consent Form.

# 9.3.4. Access to Information for Auditing or Inspections

Representatives of regulatory authorities or of Gilead may conduct inspections or audits of the clinical study. If the investigator is notified of an inspection by a regulatory authority the investigator agrees to notify the Gilead medical monitor immediately. The investigator agrees to provide to representatives of a regulatory agency or Gilead access to records, facilities, and personnel for the effective conduct of any inspection or audit.

# 9.3.5. Study Discontinuation

Both the sponsor and the investigator reserve the right to terminate the study at any time. Should this be necessary, both parties will arrange discontinuation procedures and notify the appropriate regulatory authority(ies), IRBs/IECs/ECs. In terminating the study, Gilead and the investigator will assure that adequate consideration is given to the protection of the subjects' interests.

# 10. REFERENCES

- Afzali A, Berry K, Ioannou GN. Excellent posttransplant survival for patients with nonalcoholic steatohepatitis in the United States. Liver Transpl 2012;18 (1):29-37.
- Bannas P, Kramer H, Hernando D, Agni R, Cunningham AM, Mandal R, et al. Quantitative magnetic resonance imaging of hepatic steatosis: Validation in ex vivo human livers. Hepatology 2015;62 (5):1444-55.
- Chen J, Talwalkar JA, Yin M, Glaser KJ, Sanderson SO, Ehman RL. Early detection of nonalcoholic steatohepatitis in patients with nonalcoholic fatty liver disease by using MR elastography. Radiology 2011;259 (3):749-56.
- Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron 1976:16:31-41.
- Dietrich P, Hellerbrand C. Non-alcoholic fatty liver disease, obesity and the metabolic syndrome. Best practice & research 2014;28 (4):637-53.
- Dowman JK, Tomlinson JW, Newsome PN. Pathogenesis of non-alcoholic fatty liver disease. QJM 2010;103 (2):71-83.
- Ekstedt M, Hagstrom H, Nasr P, Fredrikson M, Stal P, Kechagias S, et al. Fibrosis stage is the strongest predictor for disease-specific mortality in NAFLD after up to 33 years of follow-up [Accepted Article]. Hepatology 2014.
- Faramawi MF, Wildman RP, Gustat J, Rice J, Abdul Kareem MY. The association of the metabolic syndrome with QTc interval in NHANES III. Eur J Epidemiol 2008;23 (7):459-65.
- Kannel WB, Abbott RD, Savage DD, McNamara PM. Epidemiologic features of chronic atrial fibrillation: the Framingham study. N Engl J Med 1982;306 (17):1018-22.
- Koek GH, Liedorp PR, Bast A. The role of oxidative stress in non-alcoholic steatohepatitis. Clin Chim Acta 2011;412 (15-16):1297-305.
- Loomba R, Wolfson T, Ang B, Hooker J, Behling C, Peterson M, et al. Magnetic resonance elastography predicts advanced fibrosis in patients with nonalcoholic fatty liver disease: a prospective study. Hepatology 2014;60 (6):1920-8.
- Murakami S, Takayama F, Egashira T, Imao M, Mori A. Fermented papaya preparation halts the progression of non-alcoholic steatohepatitis in rats. Journal of Biophysical Chemisty 2013;4 (2):84-90.


- Nakamoto K, Takayama F, Mankura M, Hidaka Y, Egashira T, Ogino T, et al. Beneficial Effects of Fermented Green Tea Extract in a Rat Model of Non-alcoholic Steatohepatitis. Journal of clinical biochemistry and nutrition 2009;44 (3):239-46.
- Neuschwander-Tetri BA. Hepatic lipotoxicity and the pathogenesis of nonalcoholic steatohepatitis: the central role of nontriglyceride fatty acid metabolites. Hepatology 2010;52 (2):774-88.
- Ong JP, Younossi ZM. Epidemiology and natural history of NAFLD and NASH. Clin Liver Dis 2007;11 (1):1-16, vii.
- Patel JR, Bettencourt R, Cui JY, Salotti J, Hooker J, Bhatt A, et al. Non-invasive quantitative decline in liver fat content on MRI and histologic response in nonalcoholic steatohepatitis: A secondary analysis of MOZART trial [Abstract 913]. American Assoication for the Study of Liver Diseases (AASLD); 2015 13-17 November; San Francisco, CA. pp. 659A-60A.
- Ratziu V, Thibault V, Benhamou Y, Poynard T. Successful rescue therapy with tenofovir in a patient with hepatic decompensation and adefovir resistant HBV mutant. Comp Hepatol 2006;5:1.
- Singh S, Venkatesh SK, Loomba R, Wang Z, Sirlin C, Chen J, et al. Magnetic resonance elastography for staging liver fibrosis in non-alcoholic fatty liver disease: a diagnostic accuracy systematic review and individual participant data pooled analysis. European radiology 2016;26 (5):1431-40.
- Sumida Y, Niki E, Naito Y, Yoshikawa T. Involvement of free radicals and oxidative stress in NAFLD/NASH. Free radical research 2013;47 (11):869-80.
- Vernon G, Baranova A, Younossi ZM. Systematic review: the epidemiology and natural history of non-alcoholic fatty liver disease and non-alcoholic steatohepatitis in adults. Aliment Pharmacol Ther 2011;34 (3):274-85.
- Voulgari C, Tentolouris N, Papadogiannis D, Moyssakis I, Perrea D, Kyriaki D, et al. Increased left ventricular arrhythmogenicity in metabolic syndrome and relationship with myocardial performance, risk factors for atherosclerosis, and low-grade inflammation. Metabolism: clinical and experimental 2010;59 (2):159-65.
- Wanless IR, Lentz JS. Fatty liver hepatitis (steatohepatitis) and obesity: an autopsy study with analysis of risk factors. Hepatology 1990;12 (5):1106-10.
- Williams CD, Stengel J, Asike MI, Torres DM, Shaw J, Contreras M, et al. Prevalence of nonalcoholic fatty liver disease and nonalcoholic steatohepatitis among a largely middle-aged population utilizing ultrasound and liver biopsy: a prospective study. Gastroenterology 2011;140 (1):124-31.


Wong RJ, Cheung R, Ahmed A. Nonalcoholic steatohepatitis is the most rapidly growing indication for liver transplantation in patients with hepatocellular carcinoma in the U.S. Hepatology 2014;59 (6):2188-95.

Yeh MM, Brunt EM. Pathological features of fatty liver disease. Gastroenterology 2014;147 (4):754-64.

#### 11. **APPENDICES**

| Appendix 1. | Investigator Signature Page |
|-------------|-------------------------------------|
| Appendix 2 | Study Procedures Table for GS-US-40 |

2-1852 Appendix 2. Appendix 3. CTCAE Grading Scale for Severity of Adverse Events and Laboratory

Abnormalities

Appendix 4. Pregnancy Precautions, Definition for Female of Childbearing Potential, and

Contraceptive Requirements

# Appendix 1. Investigator Signature Page

GILEAD SCIENCES, INC. 333 LAKESIDE DRIVE FOSTER CITY, CA 94404 U.S.A.

#### STUDY ACKNOWLEDGEMENT

A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety, Tolerability, and Efficacy of GS-9674 in Subjects with Nonalcoholic Steatohepatitis (NASH)

| GS-US-402-1852 Amendme | ent 1, 03 October 2016 |
|---|---|
| This protocol has been approved by Gilead Science this approval. | es, Inc. The following signature documents |
| Name (Printed) Author O3-Oct-holo Date INVESTIGATOR STATEMENT I have read the protocol, including all appendices, and I agree that it contains all necessary details for me and my staff to conduct this study as described. I will conduct this study as outlined herein and will make a reasonable effort to complete the study within the time designated. I will provide all study personnel under my supervision copies of the protocol and access to all information provided by Gilead Sciences, Inc. I will discuss this material with them to ensure | |
| Author | |
| INVESTIGATOR | STATEMENT |
| details for me and my staff to conduct this study as<br>outlined herein and will make a reasonable effort to | described. I will conduct this study as |
| [마다] : . 이 사람들은 사람들이 없었다. 다양이 아이나 아이나 아이들이 되어 없었다. 아이는 아이는 아이는 아이는 아이는 아이는 아이는 아이를 다 아이를 다 하는데 하는데 하는데 없다. 그 사람들이 아이를 다 하는데 | I discuss this material with them to ensure |
| Principal Investigator Name (Printed) | Signature |
| Date | Site Number |

# Appendix 2. Study Procedures Table for GS-US-402-1852

| | Screening | ing Treatment | | | | | | | | Follow-Up | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| _ | Week -4<br>to Day 0 <sup>a</sup> | Baseline/<br>Day 1 | Week 1<br>± 3 days | Week 4<br>± 3 days | Week 8<br>± 3 days | Week 12<br>± 7 days | Week 16<br>± 3 days | Week 20<br>± 3 days | Week 24/ET <sup>b</sup><br>± 7 days | Follow-Up <sup>b</sup> ± 5 days | Unscheduled<br>Visit <sup>y</sup> |
| Subject Fasting <sup>c</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Written Informed<br>Consent <sup>d</sup> | X | | | | | | | | | | |
| Review<br>Inclusion/Exclusion<br>Criteria | X | X | | | | | | | | | |
| Medical History | X | | | | | | | | | | |
| QoL: General<br>Assessments (CLDQ,<br>SF-36, and WPAI) <sup>e</sup> | | X | | | | X | | | X | | |
| QoL: Pruritus<br>Assessments (VAS-<br>itch and 5D-itch) <sup>e</sup> | | X | X | X | X | X | X | X | X | | |
| Complete Physical Examination | X | | | | | | | | | | |
| Symptom Driven<br>Physical Examination <sup>f</sup> | | X | X | X | X | X | X | X | X | X | X |
| Vital Signs <sup>g</sup> | X | X | X | X | X | X | X | X | X | X | |
| Weight <sup>h</sup> | X | $X^{i}$ | X | X | X | X | X | X | X <sup>i</sup> | X | X |
| Height | X | | | | | | | | | | |

| | Screening | Treatment | | | | | | | | Follow-Up | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Week -4<br>to Day 0 <sup>a</sup> | Baseline/<br>Day 1 | Week 1<br>± 3 days | Week 4<br>± 3 days | Week 8<br>± 3 days | Week 12<br>± 7 days | Week 16<br>± 3 days | Week 20<br>± 3 days | Week 24/ET <sup>b</sup><br>± 7 days | Follow-Up <sup>b</sup><br>± 5 days | Unscheduled<br>Visit <sup>y</sup> |
| Chemistry <sup>j</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Hematology <sup>k</sup> | X | X | X | X | X | X | X | X | X | X | X |
| Coagulation Panel <sup>1</sup> | X | X | X | X | X | X | X | X | X | X | |
| Lipid Profile | | X | X | X | X | X | X | X | X | | |
| Hemoglobin A1c | X | X | | | | X | | | X | | |
| Blood for<br>Biomarkers <sup>m</sup> | X | X | X | X | | X | | | X | | |
| Single PK and PD<br>Sampling | | X <sup>n</sup> | X | X | X | X | X | X | X | | |
| HIV-1, HBV and<br>HCV Serology | X | | | | | | | | | | |
| Pregnancy Test <sup>o</sup> | X | X | | X | X | X | X | X | X | X | |
| Serum FSH <sup>p</sup> | X | | | | | | | | | | |
| Genomic Sample <sup>q</sup> | | X | | | | | | | | | |
| 12-lead ECG | X | X | | | | X | | | X | | |
| Ultrasound <sup>r</sup> | X <sup>r</sup> | | | | | | | | | | |
| FibroScan®s | | X | | | | X | | | X | | |
| MRE <sup>t</sup> | X | | | | | X | | | X | | |
| MRI-PDFF <sup>t</sup> | X | | | | | X | | | X | | |
| Urine Drug Screen <sup>u</sup> | X | | | | | | | | | | |

| 2 | Screening | Treatment | | | | | | | | Follow-Up | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Week -4<br>to Day 0a | Baseline/<br>Day 1 | Week 1<br>± 3 days | Week 4<br>± 3 days | Week 8<br>± 3 days | Week 12<br>± 7 days | Week 16<br>± 3 days | Week 20<br>± 3 days | Week 24/ET <sup>b</sup><br>± 7 days | Follow-Up <sup>b</sup><br>± 5 days | Unscheduled<br>Visit <sup>y</sup> |
| Urine Collection for (Biomarker) | | X | X | X | | X | | | Х | | |
| Stool Collection for (Biomarker) | | Х | | | | | | | Х | | |
| PPD | | a. | <u> </u> | | | | | | | | |
| Dispense GS-9674<br>and PTM GS-9674 <sup>w</sup> | | X | | X | X | X | X | X | | | |
| Concomitant<br>Medications | X | Х | X | Х | X | Х | Х | Х | Х | X | Х |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X |
| Take GS-9674/ PTM<br>GS-9674 Tablets <sup>x</sup> | | | X – Daily (Baseline/ Day 1 to Week 24) | | | | | | | | |

- a. The screening visit window may be extended under special circumstances with explicit approval of the Medical Monitor. Subjects who fail to meet eligibility criteria due to an abnormal laboratory result may undergo re-testing of the abnormal analyte during the screening window. This will be done at the discretion of the investigator and with prior approval of the Medical Monitor.
- b. Subjects discontinuing the study at any time for any reason (Early Termination ET) should complete the procedures listed for the Week 24/ET Visit AND the Follow-Up visit.
- Subjects must be in a fasted state for at least 8 hours prior to blood collection.
- d. Obtain written informed consent before initiation of any screening procedure.
- e. It is recommended that QoL assessments be completed prior to any study procedures being performed and prior to the subject seeing a health care provider. Refer to the Study Reference Binder for guidance on QoL assessment administration.
- f. The focus of a symptom driven physical examination will be determined by the investigator based on subject complaint.
- g. Vital signs include blood pressure, heart rate, respiration rate, and body temperature.
- h. Refer to the Study Reference Binder for specific instructions on how weight should be measured.
- i. During the Baseline/Day 1 and Week 24 visits, measurements of waist circumference should be performed. Refer to the Study Reference Binder for specific instructions on how these measurements are to be done.

- j. Blood chemistry will include: alanine aminotransferase (ALT), aspartate aminotransferase (AST), albumin, alkaline phosphatase, bicarbonate, blood urea nitrogen (BUN), calcium, chloride, creatinine, glucose, lactate dehydrogenase (LDH), magnesium, phosphorus, potassium, sodium, total and direct bilirubin, total protein, uric acid, gamma-glutamyl transferase (GGT). Also includes C-Peptide and Insulin for the Baseline/Day 1, Week 4, 12, and 24 visits.
- k. Hematology will include: complete blood cell count with differential (red blood cells, white blood cells, platelets, and hematocrit).
- 1. Coagulation Panel includes: PT, PTT, and INR.
- m. PPD
- n. PD sampling only at Baseline/Day 1.
- o. Females of childbearing potential only (see Appendix 4). Serum pregnancy test at Screening and Urine pregnancy test at all other visits, except Week 1.
- p. Only required for some female subjects see Appendix 4.
- g. PPD
- r. Ultrasound may be performed if necessary to confirm NAFLD.
- s. Subject should be in fasted state for Fibroscan collection. Refer to the Study Reference Binder for further details. If FibroScan<sup>®</sup> is not available at a site the test may be omitted.
- t. Subjects should be in fasted state for MRE/MRI-PDFF exams. Refer to the Study Reference Binder for further details. Subject must have confirmed NAFLD before MRE/MRI-PDFF exams are done.
- u. Drug screen for amphetamines, cocaine, and opiates (ie, heroin, morphine).
- v. PPD
- w. Study drug will be assigned via the IWRS system every 4 weeks from Baseline/Day 1 through Week 20.
- x. Subjects will self-administer the study drug at the investigative site at the conclusion of the Baseline/Day 1 and Week 24 visits.
- y. If the Unscheduled visit is performed for the sole purpose of distribution of study drug, the assessments noted for this visit do not need to be performed.

# Appendix 3. CTCAE Grading Scale for Severity of Adverse Events and Laboratory Abnormalities

http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE\_4.03\_2010-06-14\_QuickReference\_8.5x11.pdf

# Appendix 4. Pregnancy Precautions, Definition for Female of Childbearing Potential, and Contraceptive Requirements

# 1) Definitions

# a. Definition of Childbearing Potential

For the purposes of this study, a female born subject is considered of childbearing potential following the initiation of puberty (Tanner stage 2) until becoming post-menopausal, unless permanently sterile or with medically documented ovarian failure.

Women are considered to be in a postmenopausal state when they are  $\geq 54$  years of age with cessation of previously occurring menses for  $\geq 12$  months without an alternative cause. In addition, women of any age with amenorrhea of  $\geq 12$  months may also be considered postmenopausal if their follicle stimulating hormone (FSH) level is in the postmenopausal range and they are not using hormonal contraception or hormonal replacement therapy.

Permanent sterilization includes hysterectomy, bilateral oophorectomy, or bilateral salpingectomy in a female subject of any age.

# b. Definition of Male Fertility

For the purposes of this study, a male born subject is considered fertile after the initiation of puberty unless permanently sterile by bilateral orchidectomy or medical documentation.

#### 2) Contraception Requirements for Female Subjects

# a. Study Drug Effects on Pregnancy and Hormonal Contraception

GS-9674 has not yet been studied in pregnant women. In initial dose range-finding studies in pregnant mice and rabbits, there were no effects on embryofetal development other than a decrease in fetal body weights in the pregnant rabbits administered 1000 mg/kg/day. The decrease in fetal body weights are likely secondary to maternal toxicity rather than a direct effect of GS-9674. The NOEL for embryo/fetal development is 300 mg/kg/day in mice and 200 mg/kg/day in rabbits. These doses were associated with exposures that are > 50-fold higher than the anticipated human exposure at the maximum proposed human dose of 100 mg once daily.

Drug-drug interaction (DDI) data do not suggest a potential for interaction with hormones used for contraception.

Please refer to the latest version of the Investigator's Brochure for additional information.

# b. Contraception Requirements for Female Subjects of Childbearing Potential

The inclusion of female subjects of childbearing potential requires the use of highly effective contraceptive measures. They must have a negative serum pregnancy test at Screening and a negative pregnancy test on the Baseline/Day 1 visit prior to randomization. Pregnancy tests will be performed at monthly intervals thereafter. Female subjects must agree to one of the following from Screening until 30 days following the last dose of the study drug, GS-9674:

• Complete abstinence from intercourse of reproductive potential. Abstinence is an acceptable method of contraception only when it is in line with the subject's preferred and usual lifestyle.

#### Or

- Consistent and correct use of 1 of the following methods of birth control listed below.
  - Intrauterine device (IUD) with a failure rate of <1% per year
  - Tubal sterilization
  - Essure micro-insert system (provided confirmation of success 3 months after procedure)
  - Vasectomy in the male partner (provided that the partner is the sole sexual partner and had confirmation of surgical success 3 months after procedure)

#### Or

- Consistent and correct use of one hormonal method and one barrier method.
  - Barrier methods
    - Diaphragm with spermicide
    - Cervical cap with spermicide
    - Male condom (with or without spermicide)
  - Hormonal methods
    - Oral contraceptives (either combined or progesterone only)
    - Injectable progesterone
    - Implants of levonorgestrel
    - Transdermal contraceptive patch
    - Contraceptive vaginal ring

Female subjects must also refrain from egg donation and in vitro fertilization during treatment and until at least 30 days after the last dose of the study drug, GS-9674.

# 3) Contraception Requirements for Male Subjects

It is theoretically possible that a relevant systemic concentration may be achieved in a female partner from exposure of the male subject's seminal fluid. Therefore, male subjects with female partners of childbearing potential must use condoms (plus spermicide) during treatment and until 90 days after the last dose of GS-9674. Additional contraception recommendations should also be considered if the female partner is not pregnant.

Male subjects must also refrain from sperm donation during treatment and until at least 90 days after the last dose of the study drug, GS-9674.

# 4) Unacceptable Birth Control Methods

Birth control methods that are unacceptable include periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method (LAM). Female condom and male condom should not be used together.

# 5) Procedures to be Followed in the Event of Pregnancy

Subjects will be instructed to notify the investigator if they become pregnant at any time during the study, or if they become pregnant within 30 days (or 90 days for the partner of male subjects) of last study drug dose. Subjects who become pregnant or who suspect that they are pregnant during the study must report the information to the investigator and discontinue study drug immediately. Subjects whose partner has become pregnant or suspects she is pregnant during the study must report the information to the investigator. Instructions for reporting pregnancy, partner pregnancy, and pregnancy outcome are outlined in Section 7.6.2.1.